CLINICAL TRIAL: NCT01175213
Title: Long-Term Tolerability and Safety of Immune Globulin Subcutaneous (IGSC) Solution Administered Subcutaneously Following Administration of Recombinant Human Hyaluronidase (rHuPH20) in Subjects With Primary Immunodeficiency Diseases
Brief Title: Tolerability and Safety of Immune Globulin Subcutaneous Solution (IGSC) and rHuPH20 in PID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160902
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Single Person; Safety; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SC/IGSC, 10% with rHuPH20 followed by SC of IGSC, 10% (safety) (Experimental): Efficacy and safety of subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10% after SC administration of recombinant human hyaluronidase (rHuPH20) followed by Safety of SC of IGSC, 10% only (safety follow-up)
  Interventions: Biological: SC treatment with IGSC, 10% with rHuPH20 followed by SC/IGSC, 10% only (safety)
- SC/IGSC, 10% with rHuPH20 followed by IV of IGSC, 10% (safety (Experimental): Efficacy and safety of subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10% after SC administration of recombinant human hyaluronidase (rHuPH20) followed by Safety of intravenous (IV) administration of IGSC, 10% only (safety follow-up)
  Interventions: Biological: SC treatment with IGSC, 10% with rHuPH20 followed by IV/IGSC, 10% only (safety)
- IV treatment with IGSC, 10% only (Experimental): Partial efficacy (trough levels of immunoglobulin G [IgG] only) and safety of intravenous (IV) administration of IGSC, 10% only. This was for participants enrolled in the study who had anti-rHuPH20 andibody titer from study160603
  Interventions: Biological: IV treatment with IGSC, 10%

INTERVENTIONS:
Biological: SC treatment with IGSC, 10% with rHuPH20 followed by SC/IGSC, 10% only (safety) — Participants are to continue on the same doses and treatment intervals of IGSC, 10% adjusted for body weight, and rHuPH20 that were used for the last infusions in Study epoch 2 of Study 160603 (NCT00814320).
  After 3 infusions, participants are to change treatment to a 2-week interval, if agreed with participant and investigator.
  During this safety follow-up period, participants are treated with IGSC, 10% via the SC route. Treatment occurred once every week. The dose was the weekly equivalent of the most recent IV dose (adjusted per body weight) and multiplied by 1.37.
  Other Names: HYQVIA (IGSC; 10% with rHuPH20 [US]); 10% with rHuPH20 [EU]); GAMMAGARD LIQUID (IGSC; 10% [US]); KIOVIG (IGSC; 10% [EU])
  Arms: SC/IGSC, 10% with rHuPH20 followed by SC of IGSC, 10% (safety)
Biological: SC treatment with IGSC, 10% with rHuPH20 followed by IV/IGSC, 10% only (safety) — Participants are to continue on the same doses and treatment intervals of IGSC, 10% adjusted for body weight, and rHuPH20 that were used for the last infusions in Study epoch 2 of Study 160603 (NCT00814320).
  After 3 infusions, participants are to change treatment to a 2-week interval, if agreed with participant and investigator.
  During this safety follow-up period, participants are treated with IGSC, 10% via the intravenous (IV) route. Treatment occurred once every 3-4 weeks. The weekly dose equivalent was 100% of the most recent IV dose.
  Other Names: GAMMAGARD LIQUID (IGSC; 10% [US]); KIOVIG (IGSC; 10% [EU]); HyQvia (IGSC; 10% with rHuPH20 [EU]); 10% with rHuPH20 [US])
  Arms: SC/IGSC, 10% with rHuPH20 followed by IV of IGSC, 10% (safety
Biological: IV treatment with IGSC, 10% — During this safety follow-up period, participants are treated with IGSC, 10% via the intravenous (IV) route.
  Other Names: GAMMAGARD LIQUID (US); KIOVIG (EU)
  Arms: IV treatment with IGSC, 10% only

SUMMARY:
The original purpose of the study is to assess the long-term safety, tolerability, and practicability of the subcutaneous (SC) treatment with Immune Globulin Subcutaneous Solution (IGSC), 10% facilitated with recombinant human hyaluronidase (rHuPH20) in participants with Primary Immunodeficiency Diseases (PID) who have completed Baxter Clinical Study Protocol No. 160603.

Following a discussion with the FDA, all participants still active in the study stopped treatment with rHuPH20 to assure safety of the participants participating in the study and went into a safety follow-up.

During this safety follow-up period, participants underwent either intravenous (IV) or SC treatment with IGSC, 10%. The IV or SC administration route was at the discretion of the participant and the investigator.

DETAILED DESCRIPTION:
IGSC, 10% is the same product as IMMUNE GLOBULIN INTRAVENOUS (HUMAN), 10% (IGIV, 10%) quoted in study 160603.

IGSC, 10% is abbreviated to IGI, 10% [IMMUNE GLOBULIN INFUSION (HUMAN), 10%]

In the US the product is licensed (trade name GAMMAGARD LIQUID) for the intravenous (IV) and SC replacement therapy of antibody deficiency in patients with PID.

In the EU this product is licensed (trade name KIOVIG)

IGSC, 10% with rHuPH20 established name is Innume Glubulin Infusion 10% (Human) with Recombinant Human Hyualuronidase.

US trade name is HYQVIA EU trade name is HyQvia

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed or is about to complete Baxter Clinical Study Protocol No. 160603. Participants who have discontinued rHuPH20 and reverted to intravenous or subcutaneous treatment due to an anti-rHuPH20 antibody also may enroll for long-term safety monitoring.
* Participant/caretaker has reviewed, signed and dated informed consent
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Participant has a serious medical condition such that the participant's safety or medical care would be impacted by participation in Study 160902
* Participant is scheduled to participate in another non-Baxter clinical study involving an investigational product or investigational device during the course of this study
* If female of childbearing potential, participant is pregnant or has a negative pregnancy test and does not agree to employ adequate birth control measures for the duration of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2013-08-06 (Actual); Study Completion 2013-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (11):
  - Cypress, California
  - Irvine, California
  - Los Angeles, California
  - San Francisco, California
  - Centennial, Colorado
  - North Palm Beach, Florida
  - Atlanta, Georgia
  - Hinsdale, Illinois
  - The Bronx, New York
  - Dallas, Texas
  - Galveston, Texas

REFERENCES:
- [Result] Wasserman RL, Melamed I, Stein MR, Engl W, Sharkhawy M, Leibl H, Puck J, Rubinstein A, Kobrynski L, Gupta S, Grant AJ, Ratnayake A, Richmond WG, Church J, Yel L, Gelmont D. Long-Term Tolerability, Safety, and Efficacy of Recombinant Human Hyaluronidase-Facilitated Subcutaneous Infusion of Human Immunoglobulin for Primary Immunodeficiency. J Clin Immunol. 2016 Aug;36(6):571-82. doi: 10.1007/s10875-016-0298-x. Epub 2016 May 25. PMID 27220317
- [Derived] Wasserman RL, Gupta S, Stein M, Rabbat CJ, Engl W, Leibl H, Yel L. Infection rates and tolerability of three different immunoglobulin administration modalities in patients with primary immunodeficiency diseases. Immunotherapy. 2022 Mar;14(4):215-224. doi: 10.2217/imt-2021-0256. Epub 2021 Dec 21. PMID 34931880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted 11 clinical sites in the United States.
Pre-assignment Details: 66 participants who enrolled from study 160603 were screened and all were enrolled on the study. Of these, 3 participants were treated with intravenous administration of Immune Globulin Intravenous (Human) (IGIV), 10% only i.e. did not receive rHuPH20 during this study.
Groups:
- IGSC - rHuPH20 Then IGSC, 10% or IGIV, 10% Only: Efficacy and safety of subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10% after SC administration of recombinant human hyaluronidase (rHuPH20). Participants then went into a safety follow-up with either SC administration of IGSC, 10% or intravenous (IV) administration of Immune Globulin Intravenous (Human) (IGIV), 10%, only. The IV or SC administration route was at the discretion of the participant and the investigator. Note: IGIV, 10% is the same product as IGSC, 10%.
- IGIV, 10% Only: Participants were treated with Immune Globulin Intravenous (Human) (IGIV), 10% only, via the intravenous (IV) route throughout the study. Note: IGIV, 10% is the same product as IGSC, 10%.
Period: IGSC, 10%/rHuPH20
Arm/Group | IGSC - rHuPH20 Then IGSC, 10% or IGIV, 10% Only | IGIV, 10% Only
Started | 63 | 3 (3 participants treated IV with IGIV,10% without rHuPH20 throughout the study.)
Completed | 48 | 3
Not Completed | 15 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Death | 1 | 0
Not completed — bone marrow transplant | 1 | 0
Not completed — clinical site closed by sponsor | 6 | 0
Not completed — site elected to exit study | 3 | 0
Period: Safety Follow-up
Arm/Group | IGSC - rHuPH20 Then IGSC, 10% or IGIV, 10% Only | IGIV, 10% Only
Started | 48 | 3
Completed | 47 | 3
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to <16 Years | Participants Aged 16 to <65 Years | Participants Aged 65 Years and Older | Total
Number analyzed (Participants) | 4 | 7 | 47 | 8 | 66
Age, Continuous [Median (Full Range); unit: Years] | 10.5 [9 to 11] | 15.0 [13 to 15] | 47.0 [16 to 64] | 71.0 [65 to 80] | 43.0 [9 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 23 | 7 | 32
  Male | 3 | 6 | 24 | 1 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 47 | 8 | 66

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Serious Bacterial Infections
Description: The point estimate of the annual rate of validated acute serious bacterial infections (VASBIs) per participant per year was provided during subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10%, after SC administration of human recombinant hyaluronidase (rHuPH20). This efficacy outcome measure was only applicable prior to the safety follow-up i.e. before discontinuation of rHuPH20.
Time Frame: Throughout the efficacy period only (from 60 to 729 days)
Population: Safety Analysis Set excluding the 3 participants who were treated with intravenous (IV) administration of IGSC, 10% without rHuPH20
Measure: Number; unit: Estimated infections/year
Groups:
- All Participants Treated With IGSC, 10% and rHuPH20: Participants treated with at least one dose of subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10% after SC administration of recombinant human hyaluronidase (rHuPH20). This does not include the 3 participants who received intravenous (IV) administration of IGSC, 10% without rHuPH20.
Arm/Group | All Participants Treated With IGSC, 10% and rHuPH20
Number analyzed (Participants) | 63
Estimated infections/year | 0.020
Statistical Analysis 1: Comparison: All Participants Treated With IGSC, 10% and rHuPH20; Test type: Superiority or Other; p < 0.0001, Poisson — Testing the null hypothesis of 1 VASBI/year against a one-sided alternative at the 0.01 level of statistical significance; Poisson = 0.020, 99% CI 1-sided [upper limit 0.045]

2. Primary Outcome: Annual Rate of All Infections
Description: Annualized rate of infections per participant as defined by MedDRA system organ class (SOC) "infections and infestations". The point estimate of the annual rate of all infections was provided during subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10%, after SC administration of human recombinant hyaluronidase (rHuPH20). This efficacy outcome measure was only applicable prior to the safety follow-up i.e. before discontinuation of rHuPH20.
Time Frame: Throughout the efficacy period only (from 60 to 729 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of infections/year
Arm/Group | All Participants Treated With IGSC, 10% and rHuPH20
Number analyzed (Participants) | 63
Number of infections/year | 2.86 [2.36 to 3.43]

3. Primary Outcome: Trough Levels of IgG Maintained During the Study Period in Relation to Dose Frequency
Description: Immunoglobulin (IgG) steady state trough levels were measured in relation to dose frequency by measuring in relation to treatment interval (2-, 3- or 4-week intervals). Initially participants were administered subcutaneous (SC) infusions of Immune Globulin Subcutaneous Solution (IGSC), 10%, after SC administration of human recombinant hyaluronidase (rHuPH20) [or IV infusions of IGSC, 10% only] at the treatment intervals and dose determined by epoch 2 of study 160603 (3- or 4-week intervals). After 3 treatment intervals (either 3- or 4- week intervals), participants changed to a 2-week treatment interval, if agreed with participant and investigator, with the dose adjusted to 1/2 of the 4-week dose or 2/3 of the 3-week dose, whichever was applicable. The rHuPH20 dose was adjusted relative to the new IGSC, 10% dose in order to achieve a dose ratio of 75 U/g IgG. This efficacy outcome measure was only applicable prior to the safety follow-up i.e. before discontinuation of rHuPH20.
Time Frame: Throughout the efficacy period only (from 60 to 729 days)
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: g/L
Groups:
- All Participants Treated With rHuPH20 and/or IGSC, 10%: All participants who had been exposed to either or both study drugs in the Safety Analysis Data Set. Study drugs are Immune Globulin Subcutaneous Solution, 10%, (IGSC, 10%) and recombinant human hyaluronidase (rHuPH20). This includes the 3 participants who received intravenous (IV) administration of IGSC, 10% without rHuPH20. The 3 participants were treated at 4-week intervals only. Number of participants in each treatment interval [N] is provided.
Arm/Group | All Participants Treated With rHuPH20 and/or IGSC, 10%
Number analyzed (Participants) | 66
g/L
  2-Week Treatment Interval [N=17] | 10.900 [9.390 to 13.300]
  3-Week Treatment Interval [N=9] | 12.300 [11.500 to 15.300]
  4-Week Treatment Interval [N=47] | 9.760 [9.260 to 10.700]

4. Secondary Outcome: The Annual Rate of Serious Adverse Events (SAEs), Related and Not Related to Study Drugs
Description: Separated into age groups as described below and into related (related to either study drug) and not related (not related to either or both study drugs). Study drugs are Immune Globulin Subcutaneous Solution (IGSC), 10% and recombinant human hyaluronidase (rHuPH20).
Time Frame: Throughout entire study period (up to 3 years). Duration of participation for each participant is variable depending on date of enrollment and their anti-rHuPH20 binding antibody titer.
Population: Safety Analysis Set
Measure: Number; unit: SAEs/year
Groups:
- IGSC, 10% - rHuPH20: Participants treated with subcutaneous (SC) administration of Immune Globulin Subcutaneous Solution (IGSC), 10% after SC administration of recombinant human hyaluronidase (rHuPH20).
- Safety Follow-up - IGSC, 10% or IGIV, 10% Only: All participants were included in the Safety Follow-up. Safety Follow-up occurred after discontinuation of treatment with recombinant human hyaluronidase (rHuPH20) and included participants who had been treated with intravenous administration of Immune Globulin Intravenous (Human) (IGIV), 10% only throughout the study (e.g. had never received rHuPH20 in this study). At Safety Follow-up, the decision for treatment with either subcutaneous (SC) administration of Immune Globulin Subcutaneous (Human) (IGSC), 10% or IV administration of IGIV, 10% was at the discretion of the investigator and participant. Note: IGIV, 10% is the same product as IGSC, 10%.
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
SAEs/year
  Participants aged 2 to <12 years - not related | 0.0000 | 0.0000
  Participants aged 2 to <12 years - related | 0.0000 | 0.0000
  Participants aged 12 to <16 years - not related | 0.0768 | 0.0000
  Participants aged 12 to <16 years - related | 0.0000 | 0.0000
  Participants aged 16 to <65 years - not related | 0.0950 | 0.0449
  Participants aged 16 to <65 years - related | 0.0000 | 0.0000
  Participants aged 65 years and older- not related | 0.5737 | 0.4728
  Participants aged 65 years and older- related | 0.0000 | 0.0000

5. Secondary Outcome: Percentage of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Interrupted or Stopped for Tolerability Concerns or for AEs
Time Frame: as for outcome 4
Population: Safety Analysis Set
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Percentage of infusions
  Percentage of infusion rates reduced | 1.3 | 0.3
  Percentage of infusions interrupted | 0.8 | 0.2
  Percentage of infusions stopped | 0.1 | 0.2

6. Secondary Outcome: Percentage of Infusions Associated With One or More Moderate or Severe AEs (Including and Excluding Infections) That Begin During or Within 72 Hours of Completion of an Infusion
Time Frame: as for outcome 4
Population: Safety Analysis Set
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Percentage of infusions
  Including Infections | 3.4 | 4.7
  Excluding Infections | 2.9 | 4.0

7. Secondary Outcome: Number of Participants Who Develop Antibodies and Neutralizing Antibodies to rHuPH20
Description: Participants who develop binding antibodies and/or neutralizing antibodies to recombinant human hyaluronidase (rHuPH20) from study 160603 and/ or from this study (160902) are included here. This study (160902) is an extension of study 160603. Study 160603 was divided into 2 study epochs. In epoch 1 of study 160603 participants were treated with intravenous (IV) administration of Immune Globulin Subcutaneous Solution (IGSC), 10%. In epoch 2 of study 160603 participants were treated with subcutaneous (SC) administration of IGSC, 10% after SC administration of rHuPH20. Only participants who completed study 160603 were eligible to be screened and enrolled in this study (160902). In this study, participants started on same doses of IGSC, 10% and rHuPH20 that were used for the last infusions in epoch 2 of study 160603.
Time Frame: Throughout entire study period for 160603 (1 year 11 months) and 160902 (2 years 11 months)
Population: Participants from study 160603 and this study (160902) who have received at least one infusion of rHuPH20
Measure: Number; unit: Number of participants
Groups:
- All Participants Treated With rHuPH20: All participants who had been exposed to recombinant human hyaluronidase (rHuPH20) in studies 160603 or 160902.
Arm/Group | All Participants Treated With rHuPH20
Number analyzed (Participants) | 66
Number of participants
  Binding antibodies (>=1:160) | 13
  Neutralizing antibodies | 0

8. Secondary Outcome: Percentage of Participants Who Develop Antibodies and Neutralizing Antibodies to rHuPH20
Description: as for outcome 7
Time Frame: Throughout entire study period for 160603 (1 year 11 months) and 160902 (2 years 11 months)
Population: Participants from study 160603 and this study (160902) who have received at least one infusion of rHuPH20
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants Treated With rHuPH20
Number analyzed (Participants) | 66
Percentage of participants
  Binding antibodies (>=1:160) | 19.7
  Neutralizing antibodies | 0

9. Secondary Outcome: Number of Participants With AEs Related to Anti-rHuPH20 Titers
Time Frame: Throughout entire study period for 160603 (1 year 11 months) and 160902 (2 years 11 months)
Population: All participants who had been exposed to recombinant human hyaluronidase (rHuPH20) in studies 160603 or 160902.
Measure: Number; unit: Number of participants
Arm/Group | All Participants Treated With rHuPH20
Number analyzed (Participants) | 13
Number of participants | 12

10. Secondary Outcome: Percentage of Participants With AEs Related to Anti-rHuPH20 Titers
Time Frame: Throughout entire study period for 160603 (1 year 11 months) and 160902 (2 years 11 months)
Population: All participants who had been exposed to recombinant human hyaluronidase (rHuPH20) in studies 160603 or 160902.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants Treated With rHuPH20
Number analyzed (Participants) | 13
Percentage of participants | 92.3

11. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to the Study Drug, and Severity (A-F).
Description: Categories presented as Preferred Term-Seriousness-Relatedness-Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relatedness to study drug: R (related to either study drug); NR (not related to either or both study drugs). Study drugs are Immune Globulin Subcutaneous Solution, 10% (IGSC, 10%) and recombinant human hyaluronidase (rHuPH20) Severity: Mild; Mod (Moderate); Severe Preferred terms abbreviated: ADHD - Attention Deficit/Hyperactivity Disorder COPD - Chronic Obstructive Pulmonary Disease Other abbreviations: CPK - Creatinine Phosphokinase Inc. - Increased Dis - Disease Sml- small
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs
  Abdominal Distension-non-SAE-R-Mild | 6 | 0
  Abdominal Hernia-non-SAE-NR-Mild | 1 | 0
  Abdominal Mass-non-SAE-NR-Mild | 0 | 1
  Abdominal Pain-non-SAE-NR-Mild | 2 | 1
  Abdominal Pain-non-SAE-NR-Mod | 4 | 0
  Abdominal Pain-non-SAE-NR-Severe | 1 | 0
  Abdominal Pain-non-SAE-R-Mild | 0 | 3
  Abdominal Pain Upper-non-SAE-NR-Mild | 7 | 0
  Abdominal Pain Upper-non-SAE-R-Mild | 1 | 0
  Abdominal Tenderness-non-SAE-NR-Mild | 2 | 0
  Abdominal Tenderness-non-SAE-R-Mild | 1 | 0
  Abnormal Loss Of Weight-non-SAE-NR-Mild | 1 | 0
  Acarodermatitis-non-SAE-NR-Mild | 2 | 1
  Acarodermatitis-non-SAE-NR-Mod | 2 | 0
  Acne-non-SAE-NR-Mild | 1 | 0
  Acne-non-SAE-NR-Mod | 1 | 0
  Actinic Keratosis-non-SAE-NR-Mild | 1 | 0
  Actinic Keratosis-non-SAE-NR-Mod | 1 | 2
  Activities of Daily Living Impaired-non-SAE-NR-Mod | 1 | 0
  Acute Sinusitis-non-SAE-NR-Mild | 0 | 1
  Acute Sinusitis-non-SAE-NR-Mod | 1 | 0
  Acute Stress Disorder-non-SAE-NR-Mild | 1 | 0
  Adhesiolysis-SAE-NR-Mod | 1 | 0
  Age Related Macular Degeneration-non-SAE-NR-Mild | 1 | 0
  Agitation-non-SAE-NR-Mild | 1 | 0
  Aldolase Increased-non-SAE-NR-Mild | 1 | 0
  Anaphylactic Reaction-non-SAE-R-Sev | 0 | 1
  Animal Bite-non-SAE-NR-Mild | 1 | 0
  Animal Scratch-non-SAE-NR-Mild | 0 | 1
  Anxiety-non-SAE-NR-Mild | 2 | 0
  Anxiety-non-SAE-NR-Mod | 2 | 0
  Aortic Calcification-non-SAE-NR-Mild | 1 | 0
  Aortic Stenosis-non-SAE-NR-Mild | 1 | 0
  Aortic Stenosis-non-SAE-NR-Mod | 1 | 0
  Aortic Valve Incompetence-non-SAE-NR-Mod | 1 | 0
  Aortic Valve Incompetence-SAE-NR-Sev | 1 | 0
  Apthous Stomatitis-non-SAE-NR-Mild | 4 | 2
  Apthous Stomatitis-non-SAE-NR-Mod | 2 | 0
  Apthous Stomatitis-non-SAE-R-Mild | 1 | 0
  Appendicitis-SAE-NR-Mod | 1 | 0
  Application Site Erythema-non-SAE-NR-Mild | 1 | 0
  Arteritis-non-SAE-NR-Mod | 1 | 0
  Arthralgia-non-SAE-NR-Mild | 7 | 1
  Arthralgia-non-SAE-NR-Mod | 0 | 6
  Arthralgia-non-SAE-R-Mild | 1 | 0
  Arthropod Bite-non-SAE-NR-Mild | 1 | 1
  Asthenia-non-SAE-NR-Mild | 1 | 0
  Asthenia-non-SAE-NR-Mod | 2 | 0
  Asthenia-non-SAE-R-Mild | 6 | 0
  Asthenia-non-SAE-R-Mod | 7 | 1
  Asthma-non-SAE-NR-Mild | 12 | 3
  Asthma-non-SAE-NR-Mod | 20 | 3
  Ataxia-non-SAE-NR-Mild | 2 | 0
  Atelectasis-non-SAE-NR-Mild | 1 | 0
  Atrial Fibrillation-non-SAE-NR-Mild | 1 | 0
  Atrial Fibrillation-SAE-NR-Mod | 1 | 0
  ADHD-non-SAE-NR-Mod | 1 | 0
  Back Pain-non-SAE-NR-Mild | 3 | 2
  Back Pain-non-SAE-NR-Mod | 3 | 2
  Back Pain-non-SAE-R-Sev | 0 | 1
  Basal Cell Carcinoma-non-SAE-NR-Mild | 1 | 0
  Basal Cell Carcinoma-non-SAE-NR-Mod | 4 | 1
  Blepharochalasis-non-SAE-NR-Mild | 1 | 0
  Blister-non-SAE-NR-Mild | 1 | 0
  Blood Bicarbonate Decreased-non-SAE-NR-Mild | 1 | 0
  Blood CPK Increased-non-SAE-NR-Mild | 3 | 0
  Blood CPK Increased-non-SAE-NR-Mod | 2 | 0
  Blood Creatinine Increased-non-SAE-NR-Mild | 1 | 0
  Blood Creatinine Increased-non-SAE-R-Mild | 0 | 1
  Blood Glucose Increased-non-SAE-NR-Mild | 4 | 1
  Blood Urea Increased-non-SAE-R-Mild | 0 | 1
  Blood Urine Present-non-SAE-NR-Mild | 2 | 0
  Body Tinea-non-SAE-NR-Mild | 2 | 0
  Bone Pain-non-SAE-NR-Mild | 1 | 0
  Breast Calcifications-non-SAE-NR-Mild | 1 | 0
  Breast Dysplasia-non-SAE-NR-Mild | 0 | 1
  Bronchiolitis-non-SAE-NR-Mild | 1 | 0
  Bronchitis-non-SAE-NR-Mild | 11 | 5
  Bronchitis-non-SAE-NR-Mod | 11 | 2
  Burns Second Degree-non-SAE-NR-Mild | 1 | 0
  Bursitis-non-SAE-NR-Mild | 2 | 0
  Candidiasis-non-SAE-NR-Mild | 1 | 0
  Cardiac Failure Congestive-SAE-NR-Mild | 1 | 0
  Cardiac Murmur-non-SAE-NR-Mod | 2 | 0
  Cardiomegaly-non-SAE-NR-Mild | 0 | 1
  Cardiomegaly-non-SAE-NR-Mod | 2 | 0
  Cardiomyopathy-non-SAE-NR-Mild | 1 | 0
  Cataract-non-SAE-NR-Mild | 1 | 1
  Cataract-non-SAE-NR-Mod | 2 | 0
  Cellulitis-non-SAE-NR-Mild | 2 | 0
  Cellulitis-non-SAE-NR-Mod | 2 | 1
  Cellulitis-SAE-NR-Mod | 0 | 1
  Cellulitis Male Ext. Genital Organ-non-SAE-NR-Mod | 1 | 0
  Cerebral Sml Vessel Ischaemic Dis-non-SAE-NR-Mild | 1 | 0
  Cerumen Impaction-non-SAE-NR-Mild | 2 | 2
  Cervical Spinal Stenosis-non-SAE-NR-Mild | 0 | 1
  Chapped Lips-non-SAE-NR-Mild | 1 | 0
  Cheilitis-non-SAE-NR-Mild | 1 | 0
  Chest Discomfort-non-SAE-NR-Mild | 1 | 0
  Chest Pain-non-SAE-NR-Mild | 2 | 0
  Chest Pain-non-SAE-NR-Mod | 1 | 0
  Chills-non-SAE-NR-Mild | 2 | 0
  Chills-non-SAE-NR-Mod | 1 | 0
  Chills-non-SAE-R-Mild | 11 | 1
  Cholelithiasis-non-SAE-NR-Mild | 2 | 0
  Chondromalacia-non-SAE-NR-Mod | 1 | 0
  Chromaturia-non-SAE-NR-Mild | 1 | 0
  COPD-non-SAE-NR-Mild | 2 | 0
  COPD-non-SAE-NR-Mod | 3 | 0
  COPD-SAE-NR-Mod | 1 | 0
  COPD-SAE-NR-Sev | 1 | 0
  Chronic Sinusitis-non-SAE-NR-Mild | 5 | 2
  Chronic Sinusitis-non-SAE-NR-Mod | 3 | 1
  Conjunctival Haemorrhage-non-SAE-NR-Mild | 1 | 0
  Conjunctival Hyperaemia-non-SAE-NR-Mild | 2 | 0
  Conjunctivitis-non-SAE-NR-Mild | 0 | 2
  Conjunctivitis Allergic-non-SAE-NR-Mild | 1 | 1
  Conjunctivitis Allergic-non-SAE-NR-Mod | 0 | 2
  Conjunctivitis Infective-non-SAE-NR-Mild | 3 | 1
  Constipation-non-SAE-NR-Mild | 3 | 3
  Constipation-non-SAE-NR-Mod | 3 | 0
  Contusion-non-SAE-NR-Mild | 0 | 3
  Convulsion-non-SAE-NR-Mild | 1 | 0
  Convulsion-non-SAE-NR-Mod | 2 | 1
  Coombs Direct Test Positive-non-SAE-R-Mild | 1 | 0
  Coombs Test Positive-non-SAE-NR-Mild | 1 | 0
  Coombs Test Positive-non-SAE-R-Mild | 1 | 0
  Corneal Abrasion-non-SAE-NR-Mild | 1 | 0
  Costochondritis-non-SAE-NR-Mild | 1 | 0
  Costochondritis-non-SAE-NR-Sev | 1 | 0
  Cough-non-SAE-NR-Mild | 10 | 3
  Cough-non-SAE-NR-Mod | 3 | 1
  Cough-non-SAE-R-Mild | 1 | 0
  Cryptosporidiosis Infection-SAE-NR-Sev | 1 | 0
  Cyst-non-SAE-NR-Mild | 1 | 0
  Cyst-non-SAE-NR-Mod | 2 | 0
  Cystitis-non-SAE-NR-Mild | 1 | 0
  Cystocele-SAE-NR-Mod | 1 | 0
  Decreased Appetite-non-SAE-NR-Mild | 1 | 0
  Decreased Appetite-non-SAE-NR-Mod | 2 | 0
  Decreased Appetite-non-SAE-R-Mild | 3 | 8
  Dehydration-non-SAE-NR-Mild | 1 | 0
  Dehydration-non-SAE-NR-Mod | 1 | 0
  Dental Caries-non-SAE-NR-Mod | 2 | 0
  Depression-non-SAE-NR-Mild | 1 | 0
  Depression-non-SAE-NR-Mod | 3 | 1
  Dermal Cyst-non-SAE-NR-Mod | 1 | 0
  Dermatitis-non-SAE-NR-Mild | 1 | 0
  Dermatitis Allergic-non-SAE-NR-Mild | 0 | 1
  Dermatitis Atopic-non-SAE-NR-Mild | 1 | 0
  Dermatitis Contact-non-SAE-NR-Mild | 3 | 0
  Dermatitis Contact-non-SAE-NR-Mod | 1 | 0
  Dermatitis Psoriasiform-non-SAE-NR-Sev | 1 | 0
  Device Breakage-non-SAE-NR-Mod | 1 | 0
  Device Failure-non-SAE-NR-Mod | 1 | 0
  Diarrhoea-non-SAE-NR-Mild | 15 | 4
  Diarrhoea-non-SAE-NR-Mod | 2 | 0
  Diarrhoea-non-SAE-R-Mild | 2 | 1
  Dizziness-non-SAE-NR-Mild | 5 | 1
  Dizziness-non-SAE-R-Mild | 5 | 0
  Dizziness-non-SAE-R-Mod | 1 | 0
  Drug Eruption-non-SAE-NR-Mod | 1 | 0
  Drug Hypersensitivity-non-SAE-NR-Mild | 3 | 0
  Dry Eye-non-SAE-NR-Mild | 1 | 0
  Dry Eye-non-SAE-NR-Mod | 1 | 1
  Dry Mouth-non-SAE-NR-Mild | 0 | 1
  Dry Skin-non-SAE-NR-Mild | 0 | 1
  Dysmenorrhoea-non-SAE-NR-Mild | 1 | 0
  Dyspepsia-non-SAE-NR-Mild | 0 | 3
  Dysplastic Naevus-non-SAE-NR-Mod | 1 | 0
  Dyspnoea-non-SAE-NR-Mild | 2 | 1
  Dyspnoea-non-SAE-NR-Mod | 2 | 0
  Dysuria-non-SAE-NR-Mild | 1 | 1
  Dysuria-non-SAE-NR-Mod | 2 | 0
  Ear Infection-non-SAE-NR-Mild | 1 | 0
  Ear Infection-non-SAE-NR-Mod | 3 | 0
  Ear Pain-non-SAE-NR-Mild | 1 | 0
  Ear Pain-non-SAE-NR-Mod | 2 | 0
  Ear Pruritus-non-SAE-R-Mild | 0 | 1
  Eccymosis-non-SAE-NR-Mild | 3 | 0
  Eccymosis-non-SAE-NR-Mod | 0 | 1
  Eczema-non-SAE-NR-Mild | 0 | 2
  Eczema-non-SAE-NR-Mod | 5 | 0
  Empty Sella Syndrome-non-SAE-NR-Mild | 1 | 0
  Epilepsy-non-SAE-NR-Mod | 1 | 0
  Epitaxis-non-SAE-NR-Mild | 11 | 5
  Erythema-non-SAE-NR-Mild | 1 | 0
  Eschar-non-SAE-NR-Mild | 1 | 0
  Excoriation-non-SAE-NR-Mild | 8 | 1
  Excoriation-non-SAE-NR-Mod | 1 | 0
  Eye Haemorrhage-non-SAE-NR-Mild | 1 | 0
  Eye Infection-non-SAE-NR-Mild | 1 | 1
  Eye Pain-non-SAE-NR-Mild | 0 | 1
  Eye Swelling-non-SAE-NR-Mild | 1 | 0
  Eyelid Ptosis-non-SAE-NR-Mild | 1 | 0
  Facial Bones Fracture-non-SAE-NR-Mod | 0 | 1
  Facial Pain-non-SAE-NR-Mod | 1 | 0
  Fall-non-SAE-NR-Mild | 3 | 1
  Fall-non-SAE-NR-Sev | 0 | 1
  Fatigue-non-SAE-NR-Mild | 7 | 1
  Fatigue-non-SAE-NR-Mod | 3 | 1
  Fatigue-non-SAE-NR-Severe | 1 | 0
  Fatigue-non-SAE-R-Mild | 13 | 14
  Fatigue-non-SAE-R-Mod | 3 | 7
  Femur Fracture-SAE-NR-Sev | 0 | 1
  Fibromyalgia-non-SAE-NR-Mod | 2 | 1
  Flatulence-non-SAE-NR-Mod | 1 | 0
  Flushing-non-SAE-NR-Mod | 1 | 0
  Folliculitis-non-SAE-NR-Mild | 1 | 0
  Food Poisoning-non-SAE-NR-Mild | 2 | 0
  Food Poisoning-non-SAE-NR-Mod | 1 | 0
  Foot Fracture-non-SAE-NR-Mod | 1 | 0
  Free Haemoglobin Present-non-SAE-NR-Mild | 1 | 0
  Free Haemoglobin Present-non-SAE-NR-Mod | 1 | 0
  Free Haemoglobin Present-non-SAE-R-Mild | 1 | 0
  Free Haemoglobin Present-non-SAE-R-Mod | 1 | 0
  Frequent Bowel Movements-non-SAE-NR-Mod | 1 | 0
  Fungal Infection-non-SAE-NR-Mild | 1 | 1
  Fungal Skin Infection-non-SAE-NR-Mild | 1 | 0

12. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to the Study Drug, and Severity (G-M).
Description: Categories presented as Preferred Term-Seriousness-Relatedness-Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relatedness to study drug: R (related to either study drug); NR (not related to either or both study drugs). Study drugs are Immune Globulin Subcutaneous Solution, 10% (IGSC, 10%) and recombinant human hyaluronidase (rHuPH20) Severity: Mild; Mod (Moderate); Severe
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs
  Gastric Stenosis-non-SAE-NR-Mod | 1 | 0
  Gastritis-non-SAE-NR-Mild | 1 | 0
  Gastroenteritis-non-SAE-NR-Mild | 3 | 0
  Gastroenteritis-non-SAE-NR-Mod | 2 | 0
  Gastroenteritis Salmonella-non-SAE-NR-Mod | 1 | 0
  Gastroenteritis Viral-non-SAE-NR-Mild | 4 | 1
  Gastroenteritis Viral-non-SAE-NR-Mod | 3 | 1
  Gastrointestinal Viral Infection-non-SAE-NR-Mild | 1 | 0
  Gastrooesophageal Reflux Disease-non-SAE-NR-Mild | 3 | 0
  Gastrooesophageal Reflux Disease-non-SAE-NR-Mod | 1 | 0
  Genital Herpes-non-SAE-NR-Mild | 2 | 2
  Genital Herpes-non-SAE-NR-Mod | 0 | 1
  Gingival Erosion-non-SAE-NR-Mild | 1 | 0
  Gingivitis-non-SAE-NR-Mild | 1 | 0
  Glaucoma-non-SAE-NR-Mod | 1 | 0
  Glycosuria-non-SAE-NR-Mild | 1 | 0
  Gout-non-SAE-NR-Mod | 1 | 0
  Haematochezia-non-SAE-NR-Mild | 1 | 0
  Haematospermia-non-SAE-NR-Mild | 1 | 0
  Haematuria-non-SAE-NR-Mild | 1 | 1
  Haemoglobin Decreased-non-SAE-R-Mild | 0 | 1
  Haemolysis-non-SAE-R-Mild | 1 | 0
  Haemorrhoids-non-SAE-NR-Mild | 2 | 0
  Haemorrhoids-non-SAE-NR-Mod | 2 | 0
  Hand Fracture-non-SAE-NR-Mod | 1 | 0
  Headache-non-SAE-NR-Mild | 22 | 5
  Headache-non-SAE-NR-Mod | 4 | 0
  Headache-non-SAE-R-Mild | 19 | 34
  Headache-non-SAE-R-Mod | 2 | 2
  Heart Rate Irregular-non-SAE-NR-Mild | 2 | 1
  Herpes Zoster-non-SAE-NR-Mod | 3 | 0
  Hiatus Hernia-non-SAE-NR-Mild | 1 | 0
  Hydrocele-non-SAE-NR-Mild | 1 | 0
  Hypercapnia-non-SAE-Mild | 1 | 0
  Hypercholesterolaemia-non-SAE-NR-Mild | 1 | 0
  Hypersensitivity-non-SAE-NR-Mild | 2 | 0
  Hypertension-non-SAE-NR-Mild | 1 | 1
  Hypertension-non-SAE-NR-Mod | 6 | 0
  Hypertension-SAE-NR-Mod | 1 | 0
  Hypoaesthesia-non-SAE-NR-Mild | 1 | 0
  Hypokalaemia-non-SAE-NR-Mild | 0 | 2
  Hypothyroidism-non-SAE-NR-Mild | 0 | 2
  Hypothyroidism-non-SAE-NR-Mod | 1 | 0
  Impetigo-non-SAE-NR-Mild | 2 | 0
  Incision Site Pain-non-SAE-NR-Mod | 1 | 0
  Increased Upper Airway Secretion-non-SAE-NR-Mild | 1 | 0
  Inflammation Of Wound-non-SAE-NR-Mild | 0 | 1
  Influenza-non-SAE-NR-Mod | 6 | 4
  Influenza Like Illness-non-SAE-NR-Mild | 3 | 0
  Influenza Like Illness-non-SAE-NR-Mod | 1 | 0
  Infusion Site Abscess-non-SAE-R-Mild | 1 | 0
  Infusion Site Bruising-non-SAE-R-Mild | 1 | 0
  Infusion Site Discolouration-non-SAE-R-Mild | 1 | 0
  Infusion Site Discomfort-non-SAE-R-Mild | 8 | 2
  Infusion Site Erythema-non-SAE-R-Mild | 22 | 0
  Infusion Site Erythema-non-SAE-R-Mod | 1 | 0
  Infusion Site Induration-non-SAE-R-Mild | 2 | 0
  Infusion Site Mass-non-SAE-R-Mild | 1 | 0
  Infusion Site Oedema-non-SAE-R-Mild | 1 | 0
  Infusion Site Pain-non-SAE-NR-Mod | 0 | 2
  Infusion Site Pain-non-SAE-R-Mild | 78 | 17
  Infusion Site Pain-non-SAE-R-Mod | 6 | 0
  Infusion Site Pruritus-non-SAE-R-Mild | 31 | 0
  Infusion Site Swelling-non-SAE-R-Mild | 3 | 0
  Infusion Site Swelling-non-SAE-R-Sev | 1 | 0
  Injection Site Pain-non-SAE-NR-Mild | 1 | 0
  Injection Site Pain-non-SAE-R-Mild | 2 | 0
  Insomnia-non-SAE-NR-Mild | 5 | 0
  Insomnia-non-SAE-NR-Mod | 0 | 1
  Intervertebral Disc Degeneration-non-SAE-NR-Mild | 1 | 0
  Iron Deficiency Anaemia-non-SAE-NR-Mild | 1 | 0
  Irritable Bowel Syndrome-non-SAE-NR-Mod | 2 | 0
  Jejunal Stenosis-non-SAE-NR-Mod | 1 | 0
  Joint Dislocation-non-SAE-NR-Sev | 1 | 0
  Joint Injury-non-SAE-NR-Mild | 2 | 0
  Joint Swelling-non-SAE-NR-Mod | 0 | 1
  Laceration-non-SAE-NR-Mild | 0 | 1
  Ligament Sprain-non-SAE-NR-Mild | 2 | 0
  Ligament Sprain-non-SAE-NR-Mod | 1 | 2
  Limb Discomfort-non-SAE-NR-Mild | 0 | 1
  Liver Function Test Abnormal-non-SAE-NR-Mild | 1 | 0
  Local Swelling-non-SAE-NR-Mild | 1 | 0
  Local Swelling-non-SAE-R-Mild | 2 | 0
  Localised Infection-non-SAE-NR-Mod | 1 | 0
  Loss Of Consciousness-non-SAE-NR-Mild | 0 | 1
  Lyme Disease-non-SAE-NR-Mild | 2 | 0
  Lymph Gland Infection-non-SAE-NR-Mod | 1 | 0
  Lymphadenitis-non-SAE-NR-Mod | 0 | 1
  Lymphadenitis Bacterial-non-SAE-NR-Mild | 2 | 0
  Lymphadenopathy-non-SAE-NR-Mild | 5 | 2
  Lymphopenia-non-SAE-NR-Mild | 1 | 0
  Malaise-non-SAE-NR-Mild | 2 | 1
  Malaise-non-SAE-R-Mild | 1 | 0
  Medical Device Pain-non-SAE-NR-Mild | 2 | 0
  Memory Impairment-non-SAE-NR-Mild | 1 | 0
  Meniscus Injury-non-SAE-NR-Mild | 1 | 0
  Menstrual Disorder-non-SAE-NR-Mod | 1 | 0
  Mental Status Changes-SAE-NR-Sev | 1 | 0
  Micturition Urgency-non-SAE-NR-Mild | 0 | 1
  Middle Ear Effusion-non-SAE-NR-Mild | 0 | 1
  Migraine-non-SAE-NR-Mild | 3 | 0
  Migraine-non-SAE-NR-Mod | 2 | 4
  Migraine-non-SAE-NR-Sev | 0 | 1
  Migraine-non-SAE-R-Mild | 1 | 2
  Migraine-non-SAE-R-Mod | 3 | 1
  Mitral Valve Incompetence-non-SAE-NR-Mild | 2 | 0
  Molluscum Contagiosum-non-SAE-NR-Mild | 1 | 1
  Mouth Ulceration-non-SAE-NR-Mild | 0 | 1
  Mucosal Inflammation-non-SAE-NR-Mild | 1 | 0
  Muscle Contractions Involuntary-non-SAE-R-Mild | 1 | 0
  Muscle Spasms-non-SAE-NR-Mild | 4 | 0
  Muscle Strain-non-SAE-NR-Mild | 2 | 0
  Muscular Weakness-non-SAE-NR-Mild | 0 | 1
  Muscular Weakness-non-SAE-NR-Mod | 1 | 0
  Musculoskeletal Pain-non-SAE-NR-Mild | 4 | 0
  Musculoskeletal Pain-non-SAE-NR-Mod | 1 | 1
  Myalgia-non-SAE-NR-Mild | 2 | 3
  Myalgia-non-SAE-NR-Mod | 0 | 1
  Myalgia-non-SAE-R-Mild | 23 | 3
  Myalgia-non-SAE-R-Mod | 3 | 1

13. Secondary Outcome: Number of All AEs Categorized by MedDRA Preferred Terms, Seriousness, Relatedness to the Study Drug, and Severity (N-Z).
Description: Categories presented as Preferred Term-Seriousness, Relatedness, Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Relatedness to study drug: R (related to either study drug); NR (not related to either or both study drugs). Study drugs are Immune Globulin Subcutaneous Solution, 10% (IGSC, 10%) and recombinant human hyaluronidase (rHuPH20) Severity: Mild; Mod (Moderate); Severe Preferred terms abbreviated: Infection - Inf.
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs
  Nasal Congestion-non-SAE-NR-Mild | 11 | 5
  Nasal Congestion-non-SAE-NR-Mod | 2 | 0
  Nasal Discomfort-non-SAE-NR-Mild | 1 | 0
  Nasopharyngitis-non-SAE-NR-Mild | 7 | 5
  Nasopharyngitis-non-SAE-NR-Mod | 1 | 0
  Nausea-non-SAE-NR-Mild | 14 | 5
  Nausea-non-SAE-NR-Mod | 4 | 1
  Nausea-non-SAE-R-Mild | 25 | 12
  Nausea-non-SAE-R-Mod | 3 | 7
  Nephrolithiasis-non-SAE-NR-Mild | 0 | 1
  Nerve Compression-non-SAE-NR-Mild | 0 | 1
  Neutrophil Count Decreased-non-SAE-NR-Mild | 0 | 1
  Ocular Hyperaemia-non-SAE-NR-Mild | 0 | 1
  Oedema Peripheral-non-SAE-NR-Mild | 4 | 4
  Oedema Peripheral-non-SAE-NR-Mod | 4 | 1
  Oedema Peripheral-non-SAE-R-Mild | 0 | 1
  Oral Candidiasis-non-SAE-NR-Mild | 2 | 0
  Oral Herpes-non-SAE-NR-Mild | 7 | 2
  Oral Pain-non-SAE-NR-Mild | 0 | 1
  Oral Pain-non-SAE-NR-Mod | 0 | 1
  Orchitis-non-SAE-NR-Mod | 1 | 0
  Oropharyngeal Pain-non-SAE-NR-Mild | 4 | 1
  Osteoarthritis-non-SAE-NR-Mild | 2 | 1
  Osteoarthritis-non-SAE-NR-Mod | 1 | 0
  Osteopenia-non-SAE-NR-Mild | 1 | 0
  Osteoporosis-non-SAE-NR-Mild | 0 | 1
  Otitis Externa-non-SAE-NR-Mild | 1 | 1
  Otitis Externa-non-SAE-NR-Mod | 0 | 1
  Otitis Media-non-SAE-NR-Mod | 1 | 1
  Pain-non-SAE-NR-Mild | 2 | 0
  Pain-non-SAE-R-Mild | 7 | 0
  Pain In Extremity-non-SAE-NR-Mild | 4 | 1
  Pain In Extremity-non-SAE-R-Sev | 0 | 1
  Palpitations-non-SAE-NR-Mild | 2 | 0
  Panic Attack-non-SAE-NR-Mild | 0 | 1
  Papule-non-SAE-NR-Mild | 1 | 0
  Paraesthesia-non-SAE-R-Mild | 1 | 0
  Paranasal Cyst-non-SAE-NR-Mild | 1 | 0
  Pelvic Pain-non-SAE-NR-Mod | 1 | 0
  Pericardial Effusion-non-SAE-NR-Mild | 1 | 0
  Perineurial Cyst-non-SAE-NR-Mod | 1 | 0
  Periodontal Disease-non-SAE-NR-Mild | 1 | 0
  Pharyngitis-non-SAE-NR-Mild | 6 | 1
  Pharyngitis-non-SAE-NR-Mod | 0 | 1
  Pharyngitis Streptococcal-non-SAE-NR-Mild | 1 | 0
  Pleural Effusion-non-SAE-NR-Mild | 1 | 0
  Pleural Effusion-non-SAE-NR-Mod | 1 | 0
  Pneumonia-non-SAE-NR-Mild | 1 | 0
  Pneumonia Bacterial-non-SAE-NR-Mod | 1 | 0
  Pneumonia Pseudomonas Aeruginosa-SAE-NR-Sev | 1 | 0
  Pollakiuria-non-SAE-NR-Mild | 0 | 1
  Pollakiuria-non-SAE-NR-Mod | 1 | 0
  Polycystic Ovaries-non-SAE-NR-Mild | 0 | 1
  Post Procedural Complication-non-SAE-NR-Mod | 1 | 0
  Post Procedural Haemorrhage-non-SAE-NR-Mild | 1 | 0
  Post Procedural Swelling-non-SAE-NR-Mild | 1 | 0
  Procedural Nausea-non-SAE-NR-Mod | 1 | 0
  Procedural Pain-non-SAE-NR-Mild | 0 | 1
  Procedural Pain-non-SAE-NR-Mod | 9 | 1
  Proctalgia-non-SAE-NR-Mod | 1 | 0
  Productive Cough-non-SAE-NR-Mild | 2 | 0
  Protein Urine Present-non-SAE-NR-Mild | 1 | 0
  Pruritus-non-SAE-NR-Mild | 3 | 3
  Pruritus-non-SAE-NR-Mod | 1 | 0
  Pruritus-non-SAE-R-Mild | 0 | 3
  Pruritus Allergic-non-SAE-NR-Mod | 0 | 1
  Pruritus Generalised-non-SAE-R-Mild | 0 | 1
  Pulmonary Hypertension-non-SAE-NR-Mild | 1 | 0
  Pulmonary Hypertension-non-SAE-NR-Mod | 1 | 0
  Pulmonary Vascular Disorder-non-SAE-NR-Mod | 1 | 0
  Puncture Site Pain-non-SAE-NR-Mild | 0 | 1
  Puncture Site Pain-non-SAE-NR-Mod | 0 | 2
  Purpura Senile-non-SAE-NR-Mild | 0 | 1
  Pyogenic Granuloma-non-SAE-NR-Mod | 1 | 1
  Pyrexia-non-SAE-NR-Mild | 11 | 5
  Pyrexia-non-SAE-NR-Mod | 2 | 0
  Pyrexia-non-SAE-R-Mild | 3 | 0
  Pyuria-non-SAE-NR-Mild | 0 | 1
  Rales-non-SAE-NR-Mod | 1 | 1
  Rash-non-SAE-NR-Mild | 2 | 1
  Rash Generalised-non-SAE-R-Mild | 0 | 1
  Rectal Polyp-non-SAE-NR-Mod | 1 | 0
  Red Blood Cells Urine Positive-non-SAE-NR-Mild | 1 | 0
  Respiratory Tract Congestion-non-SAE-NR-Mild | 2 | 0
  Respiratory Tract Congestion-non-SAE-NR-Mod | 1 | 0
  Respiratory Tract Infection-non-SAE-NR-Mild | 1 | 0
  Respiratory Tract Infection-non-SAE-NR-Mod | 1 | 0
  Restless Legs Syndrome-non-SAE-NR-Mild | 1 | 0
  Rhinitis-non-SAE-NR-Mild | 2 | 0
  Rhinitis Perennial-non-SAE-NR-Mild | 1 | 0
  Rhinorrhoea-non-SAE-NR-Mild | 2 | 1
  Rhinorrhoea-non-SAE-R-Mild | 0 | 1
  Right Atrial Dilatation-non-SAE-NR-Mild | 1 | 0
  Rotator Cuff Syndrome-non-SAE-NR-Mild | 1 | 0
  Scab-non-SAE-NR-Mild | 1 | 0
  Scar-non-SAE-NR-Mild | 1 | 0
  Scoliosis-non-SAE-NR-Mild | 0 | 1
  Scratch-non-SAE-NR-Mild | 1 | 0
  Scrotal Swelling-non-SAE-R-Mild | 3 | 0
  Seborrhoeic Keratosis-non-SAE-NR-Mod | 2 | 0
  Sinus Congestion-non-SAE-NR-Mild | 1 | 1
  Sinus Headache-non-SAE-NR-Mild | 2 | 0
  Sinusitis-non-SAE-NR-Mild | 34 | 3
  Sinusitis-non-SAE-NR-Mod | 29 | 13
  Skin Hyperpigmentation-non-SAE-NR-Mild | 1 | 0
  Skin Lesion-non-SAE-NR-Mild | 1 | 0
  Skin Mass-non-SAE-NR-Mild | 1 | 1
  Sleep Apnoea Syndrome-non-SAE-NR-Mild | 1 | 0
  Slow Speech-non-SAE-NR-Mod | 1 | 0
  Solar Lentigo-non-SAE-NR-Mild | 1 | 0
  Somnolence-non-SAE-NR-Mild | 1 | 0
  Speech Disorder-non-SAE-NR-Mild | 0 | 1
  Spermatocele-non-SAE-NR-Mild | 1 | 0
  Spinal Compression Fracture-non-SAE-NR-Mod | 1 | 0
  Spinal Meningeal Cyst-SAE-NR-Sev | 1 | 0
  Spinal Osteoarthritis-non-SAE-NR-Mild | 3 | 0
  Squamous Cell Carcinoma-non-SAE-NR-Mod | 4 | 2
  Stress-non-SAE-NR-Mod | 1 | 0
  Suicide Attempt-non-SAE-NR-Sev | 1 | 0
  Sunburn-non-SAE-NR-Mild | 1 | 0
  Swelling Face-non-SAE-NR-Mod | 1 | 0
  Swelling Face-non-SAE-NR-Sev | 0 | 1
  Swollen Tongue-non-SAE-NR-Mild | 1 | 0
  Synovial Cyst-non-SAE-NR-Mild | 1 | 0
  Tachycardia-non-SAE-NR-Mild | 5 | 1
  Tachycardia-non-SAE-Mod | 1 | 0
  Tendon Disorder-non-SAE-NR-Sev | 1 | 0
  Tendonitis-non-SAE-NR-Mild | 2 | 0
  Tendonitis-non-SAE-NR-Mod | 1 | 0
  Testicular Microlithiasis-non-SAE-NR-Mild | 1 | 0
  Testicular Pain-non-SAE-NR-Mod | 1 | 0
  Thermal Burn-non-SAE-NR-Mild | 0 | 1
  Thinking Abnormal-non-SAE-NR-Mod | 1 | 0
  Thrombocytopenia-non-SAE-NR-Mild | 1 | 0
  Tibia Fracture-non-SAE-NR-Sev | 1 | 0
  Tinea Cruris-non-SAE-NR-Mild | 1 | 0
  Tinea Infection-non-SAE-NR-Mild | 1 | 0
  Tooth Abscess-non-SAE-NR-Mild | 0 | 1
  Tooth Abscess-non-SAE-NR-Mod | 0 | 1
  Tooth Fracture-non-SAE-NR-Mod | 1 | 0
  Tooth Infection-non-SAE-NR-Mild | 1 | 0
  Tooth Infection-non-SAE-NR-Mod | 1 | 0
  Toothache-non-SAE-NR-Mod | 0 | 1
  Toxicity To Various Agents-SAE-NR-Sev | 1 | 0
  Tracheal Stenosis-non-SAE-NR-Mild | 0 | 1
  Transient Ischaemic Attack-SAE-NR-Mod | 0 | 1
  Traumatic Haematoma-non-SAE-NR-Mild | 1 | 0
  Tricuspid Valve Incompetence-non-SAE-NR-Mild | 1 | 0
  Trigeminal Neuralgia-non-SAE-NR-Mild | 1 | 0
  Tympanic Membrane Scarring-non-SAE-NR-Mild | 1 | 0
  Type 2 Diabetes Mellitus-non-SAE-NR-Mod | 2 | 0
  Upper Limb Fracture-non-SAE-NR-Mod | 1 | 0
  Upper Limb Fracture-non-SAE-NR-Sev | 1 | 0
  Upper Respiratory Tract Infection-non-SAE-NR-Mild | 16 | 8
  Upper Respiratory Tract Infection-non-SAE-NR-Mod | 13 | 2
  Upper-Airway Cough Syndrome-non-SAE-NR-Mild | 1 | 1
  Urethritis-non-SAE-NR-Mild | 1 | 0
  Urinary Tract Infection-non-SAE-NR-Mild | 4 | 4
  Urinary Tract Infection-non-SAE-NR-Mod | 6 | 2
  Urticaria-non-SAE-NR-Mild | 0 | 1
  Urticaria-non-SAE-R-Mild | 0 | 1
  Uterine Polyp-non-SAE-NR-Mod | 1 | 0
  Vaginal Prolapse-SAE-NR-Mod | 1 | 0
  Vaginitis Bacterial-non-SAE-NR-Mild | 2 | 0
  Varicose Vein-non-SAE-NR-Mild | 1 | 0
  Vasomotor Rhinitis-non-SAE-NR-Mild | 1 | 0
  Vein Pain-non-SAE-NR-Mild | 0 | 1
  Ventricular Hypokinesia-non-SAE-NR-Mild | 1 | 0
  Vessel Puncture Site Bruise-non-SAE-NR-Mild | 1 | 0
  Viral Infection-non-SAE-NR-Mild | 3 | 0
  Viral Infection-non-SAE-NR-Mod | 0 | 1
  Viral Pharyngitis-non-SAE-NR-Mild | 1 | 0
  Viral Pharyngitis-non-SAE-NR-Mod | 0 | 1
  Viral Rash-non-SAE-NR-Mod | 1 | 0
  Viral Upper Respiratory Tract Inf.-non-SAE-NR-Mild | 29 | 5
  Viral Upper Respiratory Tract Inf.-non-SAE-NR-Mod | 1 | 1
  Vision Blurred-non-SAE-NR-Mild | 1 | 0
  Vitamin B12 Deficiency-non-SAE-NR-Mild | 1 | 0
  Vitamin D Decreased-non-SAE-NR-Mild | 0 | 1
  Vitamin D Deficiency-non-SAE-NR-Mild | 2 | 0
  Vitamin D Deficiency-non-SAE-NR-Mod | 1 | 0
  Vomiting-non-SAE-NR-Mild | 13 | 2
  Vomiting-non-SAE-NR-Mod | 4 | 1
  Vomiting-non-SAE-R-Mod | 0 | 1
  Vulvar Dysplasia-non-SAE-NR-Mild | 2 | 0
  Vulvovaginal Candidiasis-non-SAE-NR-Mild | 1 | 0
  Vulvovaginal Mycotic Infection-non-SAE-NR-Mild | 4 | 1
  Vulvovaginal Mycotic Infection-non-SAE-NR-Mod | 2 | 0
  Wheezing-non-SAE-NR-Mod | 1 | 0
  Wisdom Teeth Removal-non-SAE-NR-Mild | 1 | 0
  Wisdom Teeth Removal-non-SAE-NR-Sev | 1 | 0
  Wound-non-SAE-NR-Mild | 0 | 1
  Wrist Fracture-non-SAE-NR-Mod | 0 | 1
  Xeroderma-non-SAE-NR-Mild | 1 | 0

14. Secondary Outcome: Rate of All AEs Per Participant Categorized by MedDRA Preferred Terms, Seriousness and Severity (A-F).
Description: Categories presented as Preferred Term-Seriousness-Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Severity: Mild; Mod (Moderate); Sev (Severe) Preferred terms abbreviated: ADHD - Attention Deficit/Hyperactivity Disorder COPD - Chronic Obstructive Pulmonary Disease Other abbreviations: Inc. - Increased Dis. - Disease
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs per participant
  Abdominal Distension-non-SAE-Mild | 0.095 | 0
  Abdominal Hernia-non-SAE-Mild | 0.016 | 0
  Abdominal Mass-non-SAE-Mild | 0 | 0.020
  Abdominal Pain-non-SAE-Mild | 0.032 | 0.078
  Abdominal Pain-non-SAE-Mod | 0.063 | 0
  Abdominal Pain-non-SAE-Severe | 0.016 | 0
  Abdominal Pain Upper-non-SAE-Mild | 0.127 | 0
  Abdominal Tenderness-non-SAE-Mild | 0.048 | 0
  Abnormal Loss of Weight-non-SAE-Mild | 0.016 | 0
  Acarodermatitis-non-SAE-Mild | 0.032 | 0.020
  Acarodermatitis-non-SAE-Mod | 0.032 | 0
  Acne-non-SAE-Mild | 0.016 | 0
  Acne-non-SAE-Mod | 0.016 | 0
  Actinic Keratosis-non-SAE-Mild | 0.016 | 0
  Actinic Keratosis-non-SAE-Mod | 0.016 | 0.039
  Activities of Daily Living Impaired-non-SAE-Mod | 0.016 | 0
  Acute Sinusitis-non-SAE-Mild | 0 | 0.020
  Acute Sinusitis-non-SAE-Mod | 0.016 | 0
  Acute Stress Disorder-non-SAE-Mild | 0.016 | 0
  Adhesiolysis-SAE-Mod | 0.016 | 0
  Age-Related Macular Degeneration-non-SAE-Mild | 0.016 | 0
  Agitation-non-SAE-Mild | 0.016 | 0
  Aldolase Increased-non-SAE-Mild | 0.016 | 0
  Anaphylactic Reaction-non-SAE-Sev | 0 | 0.020
  Animal Bite-non-SAE-Mild | 0.016 | 0
  Animal Scratch-non-SAE-Mild | 0 | 0.020
  Anxiety-non-SAE-Mild | 0.032 | 0
  Anxiety-non-SAE-Mod | 0.032 | 0
  Aortic Calcification-non-SAE-Mild | 0.016 | 0
  Aortic Stenosis-non-SAE-Mild | 0.016 | 0
  Aortic Stenosis-non-SAE-Mod | 0.016 | 0
  Aortic Valve Incompetence-non-SAE-Mod | 0.016 | 0
  Aortic Valve Incompetence-SAE-Sev | 0.016 | 0
  Aphthous Stomatitis-non-SAE-Mild | 0.079 | 0.039
  Aphthous Stomatitis-non-SAE-Mod | 0.032 | 0
  Appendicitis-SAE-Mod | 0.016 | 0
  Application Site Erythema-non-SAE-Mild | 0.016 | 0
  Arteritis-non-SAE-Mod | 0.016 | 0
  Arthralgia-non-SAE-Mild | 0.127 | 0.020
  Arthralgia-non-SAE-Mod | 0 | 0.118
  Arthropod Bite-non-SAE-Mild | 0.016 | 0.020
  Asthenia-non-SAE-Mild | 0.111 | 0
  Asthenia-non-SAE-Mod | 0.143 | 0.020
  Asthma-non-SAE-Mild | 0.190 | 0.059
  Asthma-non-SAE-Mod | 0.317 | 0.059
  Ataxia-non-SAE-Mild | 0.032 | 0
  Atelectasis-non-SAE-Mild | 0.016 | 0
  Atrial Fibrillation-non-SAE-Mild | 0.016 | 0
  Atrial Fibrillation-SAE-Mod | 0.016 | 0
  ADHD-non-SAE-Mod | 0.016 | 0
  Back Pain-non-SAE-Mild | 0.048 | 0.039
  Back Pain-non-SAE-Mod | 0.048 | 0.039
  Back Pain-non-SAE-Sev | 0 | 0.020
  Basal Cell Carcinoma-non-SAE-Mild | 0.016 | 0
  Basal Cell Carcinoma-non-SAE-Mod | 0.063 | 0.020
  Blepharochalasis-non-SAE-Mild | 0.016 | 0
  Blister-non-SAE-Mild | 0.016 | 0
  Blood Bicarbonate Decreased-non-SAE-Mild | 0.016 | 0
  Blood Creatine Phosphokinase Inc.-non-SAE-Mild | 0.048 | 0
  Blood Creatine Phosphokinase Inc.-non-SAE-Mod | 0.032 | 0
  Blood Creatinine Increased-non-SAE-Mild | 0.016 | 0.020
  Blood Glucose Increased-non-SAE-Mild | 0.063 | 0.020
  Blood Urea Increased-non-SAE-Mild | 0 | 0.020
  Blood Urine Present-non-SAE-Mild | 0.032 | 0
  Body Tinea-non-SAE-Mild | 0.032 | 0
  Bone Pain-non-SAE-Mild | 0.016 | 0
  Breast Calcifications-non-SAE-Mild | 0.016 | 0
  Breast Dysplasia-non-SAE-Mild | 0 | 0.020
  Bronchiolitis-non-SAE-Mild | 0.016 | 0
  Bronchitis-non-SAE-Mild | 0.175 | 0.098
  Bronchitis-non-SAE-Mod | 0.175 | 0.039
  Burns Second Degree-non-SAE-Mild | 0.016 | 0
  Bursitis-non-SAE-Mild | 0.032 | 0
  Candidiasis-non-SAE-Mild | 0.016 | 0
  Cardiac Failure Congestive-SAE-Mild | 0.016 | 0
  Cardiac Murmur-non-SAE-Mild | 0.032 | 0
  Cardiomegaly-non-SAE-Mild | 0 | 0.020
  Cardiomegaly-non-SAE-Mod | 0.032 | 0
  Cardiomyopathy-non-SAE-Mild | 0.016 | 0
  Cataract-non-SAE-Mild | 0.016 | 0.020
  Cataract-non-SAE-Mod | 0.032 | 0
  Cellulitis-non-SAE-Mild | 0.032 | 0
  Cellulitis-non-SAE-Mod | 0.032 | 0.020
  Cellulitis-SAE-Mod | 0 | 0.020
  Cellulitis Of Male Ext Genital Organ-non-SAE-Mod | 0.016 | 0
  Cerebral Small Vessel Ischaemic Dis.-non-SAE-Mild | 0.016 | 0
  Cerumen Impaction-non-SAE-Mild | 0.032 | 0.039
  Cervical Spinal Stenosis-non-SAE-Mild | 0 | 0.020
  Chapped Lips-non-SAE-Mild | 0.016 | 0
  Cheilitis-non-SAE-Mild | 0.016 | 0
  Chest Discomfort-non-SAE-Mild | 0.016 | 0
  Chest Pain-non-SAE-Mild | 0.032 | 0
  Chest Pain-non-SAE-Mod | 0.016 | 0
  Chills-non-SAE-Mild | 0.206 | 0.020
  Chills-non-SAE-Mod | 0.016 | 0
  Cholelithiasis-non-SAE-Mild | 0.032 | 0
  Chondromalacia-non-SAE-Mod | 0.016 | 0
  Chromaturia-non-SAE-Mild | 0.016 | 0
  COPD-non-SAE-Mild | 0.032 | 0
  COPD-non-SAE-Mod | 0.048 | 0
  COPD-SAE-Mod | 0.016 | 0
  COPD-SAE-Sev | 0.016 | 0
  Chronic Sinusitis-non-SAE-Mild | 0.079 | 0.039
  Chronic Sinusitis-non-SAE-Mod | 0.048 | 0.020
  Conjunctival Haemorrhage-non-SAE-Mild | 0.016 | 0
  Conjunctival Hyperaemia-non-SAE-Mild | 0.032 | 0
  Conjunctivitis-non-SAE-Mild | 0 | 0.039
  Conjunctivitis Allergic-non-SAE-Mild | 0.016 | 0.020
  Conjunctivitis Allergic-non-SAE-Mod | 0 | 0.039
  Conjunctivitis Infective-non-SAE-Mild | 0.048 | 0.020
  Constipation-non-SAE-Mild | 0.048 | 0.059
  Constipation-non-SAE-Mod | 0.048 | 0
  Contusion-non-SAE-Mild | 0 | 0.059
  Convulsion-non-SAE-Mild | 0.016 | 0
  Convulsion-non-SAE-Mod | 0.032 | 0.020
  Coombs Direct Test Positive-non-SAE-Mild | 0.016 | 0
  Coombs Test Positive-non-SAE-Mild | 0.032 | 0
  Corneal Abrasion-non-SAE-Mild | 0.016 | 0
  Costochondritis-non-SAE-Mild | 0.016 | 0
  Costochondritis-non-SAE-Sev | 0.016 | 0
  Cough-non-SAE-Mild | 0.175 | 0.059
  Cough-non-SAE-Mod | 0.048 | 0.020
  Cryptosporidiosis Infection-SAE-Sev | 0.016 | 0
  Cyst-non-SAE-Mild | 0.016 | 0
  Cyst-non-SAE-Mod | 0.032 | 0
  Cystitis-non-SAE-Mild | 0.016 | 0
  Cystocele-SAE-Mod | 0.016 | 0
  Decreased Appetite-non-SAE-Mild | 0.063 | 0.157
  Decreased Appetite-non-SAE-Mod | 0.032 | 0
  Dehydration-non-SAE-Mild | 0.016 | 0
  Dehydration-non-SAE-Mod | 0.016 | 0
  Dental Caries-non-SAE-Mild | 0.032 | 0
  Depression-non-SAE-Mild | 0.016 | 0
  Depression-non-SAE-Mod | 0.048 | 0.020
  Dermal Cyst-non-SAE-Mod | 0.016 | 0
  Dermatitis-non-SAE-Mild | 0.016 | 0
  Dermatitis Allergic-non-SAE-Mild | 0 | 0.020
  Dermatitis Atopic-non-SAE-Mild | 0.016 | 0
  Dermatitis Contact-non-SAE-Mild | 0.048 | 0
  Dermatitis Contact-non-SAE-Mod | 0.016 | 0
  Dermatitis Psoriasiform-non-SAE-Sev | 0.016 | 0
  Device Breakage-non-SAE-Mod | 0.016 | 0
  Device Failure-non-SAE-Mod | 0.016 | 0
  Diarrhoea-non-SAE-Mild | 0.270 | 0.098
  Diarrhoea-non-SAE-Mod | 0.032 | 0
  Dizziness-non-SAE-Mild | 0.159 | 0.020
  Dizziness-non-SAE-Mod | 0.016 | 0
  Drug Eruption-non-SAE-Mod | 0 | 0.020
  Drug Hypersensitivity-non-SAE-Mild | 0.048 | 0
  Dry Eye-non-SAE-Mild | 0.016 | 0
  Dry Eye-non-SAE-Mod | 0.016 | 0.020
  Dry Mouth-non-SAE-Mild | 0 | 0.020
  Dry Skin-non-SAE-Mild | 0 | 0.020
  Dysmenorrhoea-non-SAE-Mild | 0.016 | 0
  Dyspepsia-non-SAE-Mild | 0 | 0.059
  Dysplastic Naevus-non-SAE-Mod | 0.016 | 0
  Dyspnoea-non-SAE-Mild | 0.032 | 0.020
  Dyspnoea-non-SAE-Mod | 0.032 | 0
  Dysuria-non-SAE-Mild | 0.016 | 0.020
  Dysuria-non-SAE-Mod | 0.032 | 0
  Ear Infection-non-SAE-Mild | 0.016 | 0
  Ear Infection-non-SAE-Mod | 0.048 | 0
  Ear Pain-non-SAE-Mild | 0.016 | 0
  Ear Pain-non-SAE-Mod | 0.032 | 0
  Ear Pruritus-non-SAE-Mild | 0 | 0.020
  Ecchymosis-non-SAE-Mild | 0.048 | 0
  Ecchymosis-non-SAE-Mod | 0 | 0.020
  Eczema-non-SAE-Mild | 0 | 0.039
  Eczema-non-SAE-Mod | 0.079 | 0
  Empty Sella Syndrome-non-SAE-Mild | 0.016 | 0
  Epilepsy-non-SAE-Mod | 0.016 | 0
  Epistaxis-non-SAE-Mild | 0.175 | 0.098
  Erythema-non-SAE-Mild | 0.016 | 0
  Eschar-non-SAE-Mild | 0.016 | 0
  Excoriation-non-SAE-Mild | 0.127 | 0.020
  Excoriation-non-SAE-Mod | 0.016 | 0
  Eye Haemorrhage-non-SAE-Mild | 0.016 | 0
  Eye Infection-non-SAE-Mild | 0.016 | 0.020
  Eye Pain-non-SAE-Mild | 0 | 0.020
  Eye Swelling-non-SAE-Mild | 0.016 | 0
  Eyelid Ptosis-non-SAE-Mild | 0.016 | 0
  Facial Bones Fracture-non-SAE-Mod | 0 | 0.020
  Facial Pain-non-SAE-Mod | 0.016 | 0
  Fall-non-SAE-Mild | 0.048 | 0.020
  Fall-non-SAE-Sev | 0 | 0.020
  Fatigue-non-SAE-Mild | 0.317 | 0.294
  Fatigue-non-SAE-Mod | 0.095 | 0.157
  Fatigue-non-SAE-Sev | 0.016 | 0
  Femur Fracture-SAE-Sev | 0 | 0.020
  Fibromyalgia-non-SAE-Mod | 0.032 | 0.020
  Flatulence-non-SAE-Mod | 0.016 | 0
  Flushing-non-SAE-Mod | 0 | 0.020
  Folliculitis-non-SAE-Mild | 0.016 | 0
  Food Poisoning-non-SAE-Mild | 0.032 | 0
  Food Poisoning-non-SAE-Mod | 0.016 | 0
  Foot Fracture-non-SAE-Mod | 0.016 | 0
  Free Haemoglobin Present-non-SAE-Mild | 0.032 | 0
  Free Haemoglobin Present-non-SAE-Mod | 0.032 | 0
  Frequent Bowel Movements-non-SAE-Mod | 0.016 | 0
  Fungal Infection-non-SAE-Mild | 0.016 | 0.020
  Fungal Skin Infection-non-SAE-Mild | 0.016 | 0

15. Secondary Outcome: Rate of All AEs Per Participant Categorized by MedDRA Preferred Terms, Seriousness and Severity (G-M).
Description: Categories presented as Preferred term-Seriousness-Severity. The following codes are to be used: Seriousness: non-SAE-non-serious AE; SAE-serious AE Severity: Mild; Mod (Moderate); Sev (Severe)
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs per participant
  Gastric Stenosis-non-SAE-Mod | 0.016 | 0
  Gastritis-non-SAE-Mild | 0.016 | 0
  Gastroenteritis-non-SAE-Mild | 0.048 | 0
  Gastroenteritis-non-SAE-Mod | 0.032 | 0
  Gastroenteritis Salmonella-non-SAE-Mod | 0.016 | 0
  Gastroenteritis Viral-non-SAE-Mild | 0.063 | 0.020
  Gastroenteritis Viral-non-SAE-Mod | 0.048 | 0.020
  Gastrointestinal Viral Infection-non-SAE-Mild | 0.016 | 0
  Gastrooesophageal Reflux Disease-non-SAE-Mild | 0.048 | 0
  Gastrooesophageal Reflux Disease-non-SAE-Mod | 0.016 | 0
  Genital Herpes-non-SAE-Mild | 0.032 | 0.039
  Genital Herpes-non-SAE-Mod | 0 | 0.020
  Gingival Erosion-non-SAE-Mild | 0.016 | 0
  Gingivitis-non-SAE-Mild | 0.016 | 0
  Glaucoma-non-SAE-Mod | 0.016 | 0
  Glycosuria-non-SAE-Mild | 0.016 | 0
  Gout-non-SAE-Mod | 0.016 | 0
  Haematochezia-non-SAE-Mild | 0.016 | 0
  Haematospermia-non-SAE-Mild | 0.016 | 0
  Haematuria-non-SAE-Mild | 0.016 | 0.020
  Haemoglobin Decreased-non-SAE-Mild | 0 | 0.020
  Haemolysis-non-SAE-Mild | 0.016 | 0
  Haemorrhoids-non-SAE-Mild | 0.032 | 0
  Haemorrhoids-non-SAE-Mod | 0.032 | 0
  Hand Fracture-non-SAE-Mod | 0.016 | 0
  Headache-non-SAE-Mild | 0.651 | 0.765
  Headache-non-SAE-Mod | 0.095 | 0.039
  Heart Rate Irregular-non-SAE-Mild | 0.032 | 0.020
  Herpes Zoster-non-SAE-Mod | 0.048 | 0
  Hiatus Hernia-non-SAE-Mild | 0.016 | 0
  Hydrocele-non-SAE-Mild | 0.016 | 0
  Hypercapnia-non-SAE-Mild | 0.016 | 0
  Hypercholesterolaemia-non-SAE-Mild | 0.016 | 0
  Hypersensitivity-non-SAE-Mild | 0.032 | 0
  Hypertension-non-SAE-Mild | 0.016 | 0.020
  Hypertension-non-SAE-Mod | 0.095 | 0
  Hypertension-SAE-Mod | 0.016 | 0
  Hypoaesthesia-non-SAE-Mild | 0.016 | 0
  Hypokalaemia-non-SAE-Mild | 0 | 0.039
  Hypothyroidism-non-SAE-Mild | 0 | 0.039
  Hypothyroidism-non-SAE-Mod | 0.016 | 0
  Impetigo-non-SAE-Mild | 0.032 | 0
  Incision Site Pain-non-SAE-Mod | 0.016 | 0
  Increased Upper Airway Secretion-non-SAE-Mild | 0.016 | 0
  Inflammation Of Wound-non-SAE-Mild | 0 | 0.020
  Influenza-non-SAE-Mod | 0.095 | 0.078
  Influenza Like Illness-non-SAE-Mild | 0.048 | 0
  Influenza Like Illness-non-SAE-Mod | 0.016 | 0
  Infusion Site Abscess-non-SAE-Mild | 0.016 | 0
  Infusion Site Bruising-non-SAE-Mild | 0.016 | 0
  Infusion Site Discolouration-non-SAE-Mild | 0.016 | 0
  Infusion Site Discomfort-non-SAE-Mild | 0.127 | 0.039
  Infusion Site Erythema-non-SAE-Mild | 0.349 | 0
  Infusion Site Erythema-non-SAE-Mod | 0.016 | 0
  Infusion Site Induration-non-SAE-Mild | 0.032 | 0
  Infusion Site Mass-non-SAE-Mild | 0.016 | 0
  Infusion Site Oedema-non-SAE-Mild | 0.016 | 0
  Infusion Site Pain-non-SAE-Mild | 1.238 | 0.333
  Infusion Site Pain-non-SAE-Mod | 0.095 | 0.039
  Infusion Site Pruritus-non-SAE-Mild | 0.492 | 0
  Infusion Site Swelling-non-SAE-Mild | 0.048 | 0
  Infusion Site Swelling-non-SAE-Sev | 0.016 | 0
  Injection Site Pain-non-SAE-Mild | 0.048 | 0
  Insomnia-non-SAE-Mild | 0.079 | 0
  Insomnia-non-SAE-Mod | 0 | 0.020
  Intervertebral Disc Degeneration-non-SAE-Mild | 0.016 | 0
  Iron Deficiency Anaemia-non-SAE-Mild | 0.016 | 0
  Irritable Bowel Syndrome-non-SAE-Mod | 0.032 | 0
  Jejunal Stenosis-non-SAE-Mod | 0.016 | 0
  Joint Dislocation-non-SAE-Sev | 0.016 | 0
  Joint Injury-non-SAE-Mild | 0.032 | 0
  Joint Swelling-non-SAE-Mod | 0 | 0.020
  Laceration-non-SAE-Mild | 0 | 0.020
  Ligament Sprain-non-SAE-Mild | 0.032 | 0
  Ligament Sprain-non-SAE-Mod | 0.016 | 0.039
  Limb Discomfort-non-SAE-Mild | 0 | 0.020
  Liver Function Test Abnormal-non-SAE-Mild | 0.016 | 0
  Local Swelling-non-SAE-Mild | 0.048 | 0
  Localised Infection-non-SAE-Mod | 0.016 | 0
  Loss Of Consciousness-non-SAE-Mild | 0 | 0.020
  Lyme Disease-non-SAE-Mild | 0.032 | 0
  Lymph Gland Infection-non-SAE-Mod | 0.016 | 0
  Lymphadenitis-non-SAE-Mod | 0 | 0.020
  Lymphadenitis Bacterial-non-SAE-Mild | 0.032 | 0
  Lymphadenopathy-non-SAE-Mild | 0.079 | 0.039
  Lymphopenia-non-SAE-Mild | 0.016 | 0
  Malaise-non-SAE-Mild | 0.048 | 0.020
  Medical Device Pain-non-SAE-Mild | 0.032 | 0
  Memory Impairment-non-SAE-Mild | 0.016 | 0
  Meniscus Injury-non-SAE-Mild | 0.016 | 0
  Menstrual Disorder-non-SAE-Mod | 0.016 | 0
  Mental Status Changes-SAE-Sev | 0.016 | 0
  Micturition Urgency-non-SAE-Mild | 0 | 0.020
  Middle Ear Effusion-non-SAE-Mild | 0 | 0.020
  Migraine-non-SAE-Mild | 0.063 | 0.039
  Migraine-non-SAE-Mod | 0.079 | 0.098
  Migraine-non-SAE-Sev | 0 | 0.020
  Mitral Valve Incompetence-non-SAE-Mild | 0.032 | 0
  Molluscum Contagiosum-non-SAE-Mild | 0.016 | 0.020
  Mouth Ulceration-non-SAE-Mild | 0 | 0.020
  Mucosal Inflammation-non-SAE-Mild | 0.016 | 0
  Muscle Contractions Involuntary-non-SAE-Mild | 0.016 | 0
  Muscle Spasms-non-SAE-Mild | 0.063 | 0
  Muscle Strain-non-SAE-Mild | 0.032 | 0
  Muscular Weakness-non-SAE-Mild | 0 | 0.020
  Muscular Weakness-non-SAE-Mod | 0.016 | 0
  Musculoskeletal Pain-non-SAE-Mild | 0.063 | 0
  Musculoskeletal Pain-non-SAE-Mod | 0.016 | 0.020
  Myalgia-non-SAE-Mild | 0.397 | 0.118
  Myalgia-non-SAE-Mod | 0.048 | 0.039

16. Secondary Outcome: Rate of All AEs Per Participant Categorized by MedDRA Preferred Terms, Seriousness and Severity (N-Z).
Description: as for outcome 15
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs per participant
  Nasal Congestion-non-SAE-Mild | 0.175 | 0.098
  Nasal Congestion-non-SAE-Mod | 0.032 | 0
  Nasal Discomfort-non-SAE-Mild | 0.016 | 0
  Nasopharyngitis-non-SAE-Mild | 0.111 | 0.098
  Nasopharyngitis-non-SAE-Mod | 0.016 | 0
  Nausea-non-SAE-Mild | 0.619 | 0.333
  Nausea-non-SAE-Mod | 0.111 | 0.157
  Nephrolithiasis-non-SAE-Mild | 0 | 0.020
  Nerve Compression-non-SAE-Mild | 0 | 0.020
  Neutrophil Count Decreased-non-SAE-Mild | 0 | 0.020
  Ocular Hyperaemia-non-SAE-Mild | 0 | 0.020
  Oedema Peripheral-non-SAE-Mild | 0.063 | 0.098
  Oedema Peripheral-non-SAE-Mod | 0.063 | 0.020
  Oral Candidiasis-non-SAE-Mild | 0.032 | 0
  Oral Herpes-non-SAE-Mild | 0.111 | 0.039
  Oral Pain-non-SAE-Mild | 0 | 0.020
  Oral Pain-non-SAE-Mod | 0 | 0.020
  Orchitis-non-SAE-Mod | 0.016 | 0
  Oropharyngeal Pain-non-SAE-Mild | 0.063 | 0.020
  Osteoarthritis-non-SAE-Mild | 0.032 | 0.020
  Osteoarthritis-non-SAE-Mod | 0.016 | 0
  Osteopenia-non-SAE-Mild | 0.016 | 0
  Osteoporosis-non-SAE-Mild | 0 | 0.020
  Otitis Externa-non-SAE-Mild | 0.016 | 0.020
  Otitis Externa-non-SAE-Mod | 0 | 0.020
  Otitis Media-non-SAE-Mod | 0.016 | 0.020
  Pain-non-SAE-Mild | 0.143 | 0
  Pain In Extremity-non-SAE-Mild | 0.063 | 0.020
  Pain In Extremity-non-SAE-Sev | 0 | 0.020
  Palpitations-non-SAE-Mild | 0.032 | 0
  Panic Attack-non-SAE-Mild | 0 | 0.020
  Papule-non-SAE-Mild | 0.016 | 0
  Paraesthesia-non-SAE-Mild | 0.016 | 0
  Paranasal Cyst-non-SAE-Mild | 0.016 | 0
  Pelvic Pain-non-SAE-Mod | 0.016 | 0
  Pericardial Effusion-non-SAE-Mild | 0.016 | 0
  Perineurial Cyst-non-SAE-Mod | 0.016 | 0
  Periodontal Disease-non-SAE-Mild | 0.016 | 0
  Pharyngitis-non-SAE-Mild | 0.095 | 0.020
  Pharyngitis-non-SAE-Mod | 0 | 0.020
  Pharyngitis Streptococcal-non-SAE-Mild | 0.016 | 0
  Pleural Effusion-non-SAE-Mild | 0.016 | 0
  Pleural Effusion-non-SAE-Mod | 0.016 | 0
  Pneumonia-non-SAE-Mild | 0.016 | 0
  Pneumonia Bacterial-non-SAE-Mod | 0.016 | 0
  Pneumonia Pseudomonas Aeruginosa-SAE-Sev | 0.016 | 0
  Pollakiuria-non-SAE-Mild | 0 | 0.020
  Pollakiuria-non-SAE-Mod | 0.016 | 0
  Polycystic Ovaries-non-SAE-Mild | 0 | 0.020
  Post Procedural Complication-non-SAE-Mod | 0.016 | 0
  Post Procedural Haemorrhage-non-SAE-Mild | 0.016 | 0
  Post Procedural Swelling-non-SAE-Mild | 0.016 | 0
  Procedural Nausea-non-SAE-Mod | 0.016 | 0
  Procedural Pain-non-SAE-Mild | 0 | 0.020
  Procedural Pain-non-SAE-Mod | 0.143 | 0.020
  Proctalgia-non-SAE-Mod | 0.016 | 0
  Productive Cough-non-SAE-Mild | 0.032 | 0
  Protein Urine Present-non-SAE-Mild | 0.016 | 0
  Pruritus-non-SAE-Mild | 0.048 | 0.118
  Pruritus-non-SAE-Mod | 0.016 | 0
  Pruritus Allergic-non-SAE-Mod | 0 | 0.020
  Pruritus Generalised-non-SAE-Mild | 0 | 0.020
  Pulmonary Hypertension-non-SAE-Mild | 0.016 | 0
  Pulmonary Hypertension-non-SAE-Mod | 0.016 | 0
  Pulmonary Vascular Disorder-non-SAE-Mod | 0.016 | 0
  Puncture Site Pain-non-SAE-Mild | 0 | 0.020
  Puncture Site Pain-non-SAE-Mod | 0 | 0.039
  Purpura Senile-non-SAE-Mild | 0 | 0.020
  Pyogenic Granuloma-non-SAE-Mod | 0.016 | 0.020
  Pyrexia-non-SAE-Mild | 0.222 | 0.098
  Pyrexia-non-SAE-Mod | 0.032 | 0
  Pyuria-non-SAE-Mild | 0 | 0.020
  Rales-non-SAE-Mod | 0.016 | 0.020
  Rash-non-SAE-Mild | 0.032 | 0.020
  Rash Generalised-non-SAE-Mild | 0 | 0.020
  Rectal Polyp-non-SAE-Mod | 0.016 | 0
  Red Blood Cells Urine Positive-non-SAE-Mild | 0.016 | 0
  Respiratory Tract Congestion-non-SAE-Mild | 0.032 | 0
  Respiratory Tract Congestion-non-SAE-Mod | 0.016 | 0
  Respiratory Tract Infection-non-SAE-Mild | 0.016 | 0
  Respiratory Tract Infection-non-SAE-Mod | 0.016 | 0
  Restless Legs Syndrome-non-SAE-Mild | 0.016 | 0
  Rhinitis-non-SAE-Mild | 0.032 | 0
  Rhinitis Perennial-non-SAE-Mild | 0.016 | 0
  Rhinorrhoea-non-SAE-Mild | 0.032 | 0.039
  Right Atrial Dilatation-non-SAE-Mild | 0.016 | 0
  Rotator Cuff Syndrome-non-SAE-Mild | 0.016 | 0
  Scab-non-SAE-Mild | 0.016 | 0
  Scar-non-SAE-Mild | 0.016 | 0
  Scoliosis-non-SAE-Mild | 0 | 0.020
  Scratch-non-SAE-Mild | 0.016 | 0
  Scrotal Swelling-non-SAE-Mild | 0.048 | 0
  Seborrhoeic Keratosis-non-SAE-Mod | 0.032 | 0
  Sinus Congestion-non-SAE-Mild | 0.016 | 0.020
  Sinus Headache-non-SAE-Mild | 0.032 | 0
  Sinusitis-non-SAE-Mild | 0.540 | 0.059
  Sinusitis-non-SAE-Mod | 0.460 | 0.255
  Skin Hyperpigmentation-non-SAE-Mild | 0.016 | 0
  Skin Lesion-non-SAE-Mild | 0.016 | 0
  Skin Mass-non-SAE-Mild | 0.016 | 0.020
  Sleep Apnoea Syndrome-non-SAE-Mild | 0.016 | 0
  Slow Speech-non-SAE-Mod | 0.016 | 0
  Solar Lentigo-non-SAE-Mild | 0.016 | 0
  Somnolence-non-SAE-Mild | 0.016 | 0
  Speech Disorder-non-SAE-Mild | 0 | 0.020
  Spermatocele-non-SAE-Mild | 0.016 | 0
  Spinal Compression Fracture-non-SAE-Mod | 0.016 | 0
  Spinal Meningeal Cyst-SAE-Sev | 0.016 | 0
  Spinal Osteoarthritis-non-SAE-Mild | 0.048 | 0
  Squamous Cell Carcinoma-non-SAE-Mod | 0.063 | 0.039
  Stress-non-SAE-Mod | 0.016 | 0
  Suicide Attempt-non-SAE-Sev | 0.016 | 0
  Sunburn-non-SAE-Mild | 0.016 | 0
  Swelling Face-non-SAE-Mod | 0.016 | 0
  Swelling Face-non-SAE-Sev | 0 | 0.020
  Swollen Tongue-non-SAE-Mild | 0.016 | 0
  Synovial Cyst-non-SAE-Mild | 0.016 | 0
  Tachycardia-non-SAE-Mild | 0.079 | 0.020
  Tachycardia-non-SAE-Mod | 0.016 | 0
  Tendon Disorder-non-SAE-Sev | 0.016 | 0
  Tendonitis-non-SAE-Mild | 0.032 | 0
  Tendonitis-non-SAE-Mod | 0.016 | 0
  Testicular Microlithiasis-non-SAE-Mild | 0.016 | 0
  Testicular Pain-non-SAE-Mod | 0.016 | 0
  Thermal Burn-non-SAE-Mild | 0 | 0.020
  Thinking Abnormal-non-SAE-Mod | 0.016 | 0
  Thrombocytopenia-non-SAE-Mild | 0.016 | 0
  Tibia Fracture-non-SAE-Sev | 0.016 | 0
  Tinea Cruris-non-SAE-Mild | 0.016 | 0
  Tinea Infection-non-SAE-Mild | 0.016 | 0
  Tooth Abscess-non-SAE-Mild | 0 | 0.020
  Tooth Abscess-non-SAE-Mod | 0 | 0.020
  Tooth Fracture-non-SAE-Mod | 0.016 | 0
  Tooth Infection-non-SAE-Mild | 0.016 | 0
  Tooth Infection-non-SAE-Mod | 0.016 | 0
  Toothache-non-SAE-Mod | 0 | 0.020
  Toxicity To Various Agents-SAE-Sev | 0.016 | 0
  Tracheal Stenosis-non-SAE-Mild | 0 | 0.020
  Transient Ischaemic Attack-SAE-Mod | 0 | 0.020
  Traumatic Haematoma-non-SAE-Mild | 0.016 | 0
  Tricuspid Valve Incompetence-non-SAE-Mild | 0.016 | 0
  Trigeminal Neuralgia-non-SAE-Mild | 0.016 | 0
  Tympanic Membrane Scarring-non-SAE-Mild | 0.016 | 0
  Type 2 Diabetes Mellitus-non-SAE-Mod | 0.032 | 0
  Upper Limb Fracture-non-SAE-Mod | 0.016 | 0
  Upper Limb Fracture-non-SAE-Sev | 0.016 | 0
  Upper Respiratory Tract Infection-non-SAE-Mild | 0.254 | 0.157
  Upper Respiratory Tract Infection-non-SAE-Mod | 0.206 | 0.039
  Upper-Airway Cough Syndrome-non-SAE-Mild | 0.016 | 0.020
  Urethritis-non-SAE-Mild | 0.016 | 0
  Urinary Tract Infection-non-SAE-Mild | 0.063 | 0.078
  Urinary Tract Infection-non-SAE-Mod | 0.095 | 0.039
  Urticaria-non-SAE-Mild | 0 | 0.039
  Uterine Polyp-non-SAE-Mod | 0.016 | 0
  Vaginal Prolapse-SAE-Mod | 0.016 | 0
  Vaginitis Bacterial-non-SAE-Mild | 0.032 | 0
  Varicose Vein-non-SAE-Mild | 0.016 | 0
  Vasomotor Rhinitis-non-SAE-Mild | 0.016 | 0
  Vein Pain-non-SAE-Mild | 0 | 0.020
  Ventricular Hypokinesia-non-SAE-Mild | 0.016 | 0
  Vessel Puncture Site Bruise-non-SAE-Mild | 0.016 | 0
  Viral Infection-non-SAE-Mild | 0.048 | 0
  Viral Infection-non-SAE-Mod | 0 | 0.020
  Viral Pharyngitis-non-SAE-Mild | 0.016 | 0
  Viral Pharyngitis-non-SAE-Mod | 0 | 0.020
  Viral Rash-non-SAE-Mod | 0.016 | 0
  Viral Upper Respiratory Tract Inf.-non-SAE-Mild | 0.460 | 0.098
  Viral Upper Respiratory Tract Inf-non-SAE-Mod | 0.016 | 0.020
  Vision Blurred-non-SAE-Mild | 0.016 | 0
  Vitamin B12 Deficiency-non-SAE-Mild | 0.016 | 0
  Vitamin D Decreased-non-SAE-Mild | 0 | 0.020
  Vitamin D Deficiency-non-SAE-Mild | 0.032 | 0
  Vitamin D Deficiency-non-SAE-Mod | 0.016 | 0
  Vomiting-non-SAE-Mild | 0.206 | 0.039
  Vomiting-non-SAE-Mod | 0.063 | 0.039
  Vulvar Dysplasia-non-SAE-Mild | 0.032 | 0
  Vulvovaginal Candidiasis-non-SAE-Mild | 0.016 | 0
  Vulvovaginal Mycotic Infection-non-SAE-Mild | 0.063 | 0.020
  Vulvovaginal Mycotic Infection-non-SAE-Mod | 0.032 | 0
  Wheezing-non-SAE-Mod | 0.016 | 0
  Wisdom Teeth Removal-non-SAE-Mild | 0.016 | 0
  Wisdom Teeth Removal-non-SAE-Sev | 0.016 | 0
  Wound-non-SAE-Mild | 0 | 0.020
  Wrist Fracture-non-SAE-Mod | 0 | 0.020
  Xeroderma-non-SAE-Mild | 0.016 | 0

17. Secondary Outcome: Rate of All AEs Per Infusion Categorized by MedDRA Preferred Terms, Seriousness and Severity (A-F).
Description: Categories presented as Preferred term-Seriousness-Severity. The following codes are to be used: Seriousness: non-SAE-non-serious adverse event; SAE- serious adverse event Severity: Mild; Mod (Moderate); Sev (Severe) Preferred terms abbreviated: ADHD - Attention Deficit/Hyperactivity Disorder COPD - Chronic Obstructive Pulmonary Disease Other abbreviations: Inc. - Increased Dis. - Disease
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Number of AEs per infusion
  Abdominal Distension-non-SAE-Mild | 0.004 | 0
  Abdominal Hernia-non-SAE-Mild | 0.001 | 0
  Abdominal Mass-non-SAE-Mild | 0.002 | 0
  Abdominal Pain-non-SAE-Mild | 0.001 | 0.007
  Abdominal Pain-non-SAE-Mod | 0.003 | 0
  Abdominal Pain-non-SAE-Severe | 0.001 | 0
  Abdominal Pain Upper-non-SAE-Mild | 0.005 | 0
  Abdominal Tenderness-non-SAE-Mild | 0.002 | 0
  Abnormal Loss of Weight-non-SAE-Mild | 0.001 | 0
  Acarodermatitis-non-SAE-Mild | 0.001 | 0.002
  Acarodermatitis-non-SAE-Mod | 0.001 | 0
  Acne-non-SAE-Mild | 0.001 | 0
  Acne-non-SAE-Mod | 0.001 | 0
  Actinic Keratosis-non-SAE-Mild | 0.001 | 0
  Actinic Keratosis-non-SAE-Mod | 0.001 | 0.003
  Activities of Daily Living Impaired-non-SAE-Mod | 0.001 | 0
  Acute Sinusitis-non-SAE-Mild | 0 | 0.002
  Acute Sinusitis-non-SAE-Mod | 0.001 | 0
  Acute Stress Disorder-non-SAE-Mild | 0.001 | 0
  Adhesiolysis-SAE-Mod | 0.001 | 0
  Age-Related Macular Degeneration-non-SAE-Mild | 0.001 | 0
  Agitation-non-SAE-Mild | 0.001 | 0
  Aldolase Increased-non-SAE-Mild | 0.001 | 0
  Anaphylactic Reaction-non-SAE-Sev | 0 | 0.002
  Animal Bite-non-SAE-Mild | 0.001 | 0
  Animal Scratch-non-SAE-Mild | 0 | 0.002
  Anxiety-non-SAE-Mild | 0.001 | 0
  Anxiety-non-SAE-Mod | 0.001 | 0
  Aortic Calcification-non-SAE-Mild | 0.001 | 0
  Aortic Stenosis-non-SAE-Mild | 0.001 | 0
  Aortic Stenosis-non-SAE-Mod | 0.001 | 0
  Aortic Valve Incompetence-non-SAE-Mod | 0.001 | 0
  Aortic Valve Incompetence-SAE-Sev | 0.001 | 0
  Aphthous Stomatitis-non-SAE-Mild | 0.003 | 0.003
  Aphthous Stomatitis-non-SAE-Mod | 0.001 | 0
  Appendicitis-SAE-Mod | 0.001 | 0
  Application Site Erythema-non-SAE-Mild | 0.001 | 0
  Arteritis-non-SAE-Mod | 0.001 | 0
  Arthralgia-non-SAE-Mild | 0.005 | 0.002
  Arthralgia-non-SAE-Mod | 0 | 0.010
  Arthropod Bite-non-SAE-Mild | 0.001 | 0.002
  Asthenia-non-SAE-Mild | 0.004 | 0
  Asthenia-non-SAE-Mod | 0.006 | 0.002
  Asthma-non-SAE-Mild | 0.008 | 0.005
  Asthma-non-SAE-Mod | 0.013 | 0.005
  Ataxia-non-SAE-Mild | 0.001 | 0
  Atelectasis-non-SAE-Mild | 0.001 | 0
  Atrial Fibrillation-non-SAE-Mild | 0.001 | 0
  Atrial Fibrillation-SAE-Mod | 0.001 | 0
  ADHD-non-SAE-Mod | 0.001 | 0
  Back Pain-non-SAE-Mild | 0.002 | 0.003
  Back Pain-non-SAE-Mod | 0.002 | 0.003
  Back Pain-non-SAE-Sev | 0 | 0.002
  Basal Cell Carcinoma-non-SAE-Mild | 0.001 | 0
  Basal Cell Carcinoma-non-SAE-Mod | 0.003 | 0.002
  Blepharochalasis-non-SAE-Mild | 0.001 | 0
  Blister-non-SAE-Mild | 0.001 | 0
  Blood Bicarbonate Decreased-non-SAE-Mild | 0.001 | 0
  Blood Creatine Phosphokinase Inc.-non-SAE-Mild | 0.002 | 0
  Blood Creatine Phosphokinase Inc.-non-SAE-Mod | 0.001 | 0
  Blood Creatinine Increased-non-SAE-Mild | 0.001 | 0.002
  Blood Glucose Increased-non-SAE-Mild | 0.003 | 0.002
  Blood Urea Increased-non-SAE-Mild | 0 | 0.002
  Blood Urine Present-non-SAE-Mild | 0.001 | 0
  Body Tinea-non-SAE-Mild | 0.001 | 0
  Bone Pain-non-SAE-Mild | 0.001 | 0
  Breast Calcifications-non-SAE-Mild | 0.001 | 0
  Breast Dysplasia-non-SAE-Mild | 0 | 0.002
  Bronchiolitis-non-SAE-Mild | 0.001 | 0
  Bronchitis-non-SAE-Mild | 0.007 | 0.008
  Bronchitis-non-SAE-Mod | 0.007 | 0.003
  Burns Second Degree-non-SAE-Mild | 0.001 | 0
  Bursitis-non-SAE-Mild | 0.001 | 0
  Candidiasis-non-SAE-Mild | 0.001 | 0
  Cardiac Failure Congestive-SAE-Mild | 0.001 | 0
  Cardiac Murmur-non-SAE-Mild | 0.001 | 0
  Cardiomegaly-non-SAE-Mild | 0 | 0.002
  Cardiomegaly-non-SAE-Mod | 0.001 | 0
  Cardiomyopathy-non-SAE-Mild | 0.001 | 0
  Cataract-non-SAE-Mild | 0.001 | 0.002
  Cataract-non-SAE-Mod | 0.001 | 0
  Cellulitis-non-SAE-Mild | 0.001 | 0
  Cellulitis-non-SAE-Mod | 0.001 | 0.002
  Cellulitis-SAE-Mod | 0 | 0.002
  Cellulitis Of Male Ext Genital Organ-non-SAE-Mod | 0.001 | 0
  Cerebral Small Vessel Ischaemic Dis.-non-SAE-Mild | 0.001 | 0
  Cerumen Impaction-non-SAE-Mild | 0.001 | 0.003
  Cervical Spinal Stenosis-non-SAE-Mild | 0 | 0.002
  Chapped Lips-non-SAE-Mild | 0.001 | 0
  Cheilitis-non-SAE-Mild | 0.001 | 0
  Chest Discomfort-non-SAE-Mild | 0.001 | 0
  Chest Pain-non-SAE-Mild | 0.001 | 0
  Chest Pain-non-SAE-Mod | 0.001 | 0
  Chills-non-SAE-Mild | 0.008 | 0.002
  Chills-non-SAE-Mod | 0.001 | 0
  Cholelithiasis-non-SAE-Mild | 0.001 | 0
  Chondromalacia-non-SAE-Mod | 0.001 | 0
  Chromaturia-non-SAE-Mild | 0.001 | 0
  COPD-non-SAE-Mild | 0.001 | 0
  COPD-non-SAE-Mod | 0.002 | 0
  COPD-SAE-Mod | 0.001 | 0
  COPD-SAE-Sev | 0.001 | 0
  Chronic Sinusitis-non-SAE-Mild | 0.003 | 0.003
  Chronic Sinusitis-non-SAE-Mod | 0.002 | 0.002
  Conjunctival Haemorrhage-non-SAE-Mild | 0.001 | 0
  Conjunctival Hyperaemia-non-SAE-Mild | 0.001 | 0
  Conjunctivitis-non-SAE-Mild | 0 | 0.003
  Conjunctivitis Allergic-non-SAE-Mild | 0.001 | 0.002
  Conjunctivitis Allergic-non-SAE-Mod | 0 | 0.003
  Conjunctivitis Infective-non-SAE-Mild | 0.002 | 0.002
  Constipation-non-SAE-Mild | 0.002 | 0.005
  Constipation-non-SAE-Mod | 0.002 | 0
  Contusion-non-SAE-Mild | 0 | 0.005
  Convulsion-non-SAE-Mild | 0.001 | 0
  Convulsion-non-SAE-Mod | 0.001 | 0.002
  Coombs Direct Test Positive-non-SAE-Mild | 0.001 | 0
  Coombs Test Positive-non-SAE-Mild | 0.001 | 0
  Corneal Abrasion-non-SAE-Mild | 0.001 | 0
  Costochondritis-non-SAE-Mild | 0.001 | 0
  Costochondritis-non-SAE-Sev | 0.001 | 0
  Cough-non-SAE-Mild | 0.007 | 0.005
  Cough-non-SAE-Mod | 0.002 | 0.002
  Cryptosporidiosis Infection-SAE-Sev | 0.001 | 0
  Cyst-non-SAE-Mild | 0.001 | 0
  Cyst-non-SAE-Mod | 0.001 | 0
  Cystitis-non-SAE-Mild | 0.001 | 0
  Cystocele-SAE-Mod | 0.001 | 0
  Decreased Appetite-non-SAE-Mild | 0.003 | 0.013
  Decreased Appetite-non-SAE-Mod | 0.001 | 0
  Dehydration-non-SAE-Mild | 0.001 | 0
  Dehydration-non-SAE-Mod | 0.001 | 0
  Dental Caries-non-SAE-Mild | 0.001 | 0
  Depression-non-SAE-Mild | 0.001 | 0
  Depression-non-SAE-Mod | 0.002 | 0.002
  Dermal Cyst-non-SAE-Mod | 0.001 | 0
  Dermatitis-non-SAE-Mild | 0.001 | 0
  Dermatitis Allergic-non-SAE-Mild | 0 | 0.002
  Dermatitis Atopic-non-SAE-Mild | 0.001 | 0
  Dermatitis Contact-non-SAE-Mild | 0.002 | 0
  Dermatitis Contact-non-SAE-Mod | 0.001 | 0
  Dermatitis Psoriasiform-non-SAE-Sev | 0.001 | 0
  Device Breakage-non-SAE-Mod | 0.001 | 0
  Device Failure-non-SAE-Mod | 0.001 | 0
  Diarrhoea-non-SAE-Mild | 0.011 | 0.008
  Diarrhoea-non-SAE-Mod | 0.001 | 0
  Dizziness-non-SAE-Mild | 0.006 | 0.002
  Dizziness-non-SAE-Mod | 0.001 | 0
  Drug Eruption-non-SAE-Mod | 0 | 0.002
  Drug Hypersensitivity-non-SAE-Mild | 0.002 | 0
  Dry Eye-non-SAE-Mild | 0.001 | 0
  Dry Eye-non-SAE-Mod | 0.001 | 0.002
  Dry Mouth-non-SAE-Mild | 0 | 0.002
  Dry Skin-non-SAE-Mild | 0 | 0.002
  Dysmenorrhoea-non-SAE-Mild | 0.001 | 0
  Dyspepsia-non-SAE-Mild | 0 | 0.005
  Dysplastic Naevus-non-SAE-Mod | 0.001 | 0
  Dyspnoea-non-SAE-Mild | 0.001 | 0.002
  Dyspnoea-non-SAE-Mod | 0.001 | 0
  Dysuria-non-SAE-Mild | 0.001 | 0.002
  Dysuria-non-SAE-Mod | 0.001 | 0
  Ear Infection-non-SAE-Mild | 0.001 | 0
  Ear Infection-non-SAE-Mod | 0.002 | 0
  Ear Pain-non-SAE-Mild | 0.001 | 0
  Ear Pain-non-SAE-Mod | 0.001 | 0
  Ear Pruritus-non-SAE-Mild | 0 | 0.002
  Ecchymosis-non-SAE-Mild | 0.002 | 0
  Ecchymosis-non-SAE-Mod | 0 | 0.002
  Eczema-non-SAE-Mild | 0 | 0.003
  Eczema-non-SAE-Mod | 0.003 | 0
  Empty Sella Syndrome-non-SAE-Mild | 0.001 | 0
  Epilepsy-non-SAE-Mod | 0.001 | 0
  Epistaxis-non-SAE-Mild | 0.007 | 0.008
  Erythema-non-SAE-Mild | 0.001 | 0
  Eschar-non-SAE-Mild | 0.001 | 0
  Excoriation-non-SAE-Mild | 0.005 | 0.002
  Excoriation-non-SAE-Mod | 0.001 | 0
  Eye Haemorrhage-non-SAE-Mild | 0.001 | 0
  Eye Infection-non-SAE-Mild | 0.001 | 0.002
  Eye Pain-non-SAE-Mild | 0 | 0.002
  Eye Swelling-non-SAE-Mild | 0.001 | 0
  Eyelid Ptosis-non-SAE-Mild | 0.001 | 0
  Facial Bones Fracture-non-SAE-Mod | 0 | 0.002
  Facial Pain-non-SAE-Mod | 0.001 | 0
  Fall-non-SAE-Mild | 0.002 | 0.002
  Fall-non-SAE-Sev | 0 | 0.002
  Fatigue-non-SAE-Mild | 0.013 | 0.025
  Fatigue-non-SAE-Mod | 0.004 | 0.013
  Fatigue-non-SAE-Sev | 0.001 | 0
  Femur Fracture-SAE-Sev | 0 | 0.002
  Fibromyalgia-non-SAE-Mod | 0.001 | 0.002
  Flatulence-non-SAE-Mod | 0.001 | 0
  Flushing-non-SAE-Mod | 0 | 0.002
  Folliculitis-non-SAE-Mild | 0.001 | 0
  Food Poisoning-non-SAE-Mild | 0.001 | 0
  Food Poisoning-non-SAE-Mod | 0.001 | 0
  Foot Fracture-non-SAE-Mod | 0.001 | 0
  Free Haemoglobin Present-non-SAE-Mild | 0.001 | 0
  Free Haemoglobin Present-non-SAE-Mod | 0.001 | 0
  Frequent Bowel Movements-non-SAE-Mod | 0.001 | 0
  Fungal Infection-non-SAE-Mild | 0.001 | 0.002
  Fungal Skin Infection-non-SAE-Mild | 0.001 | 0

18. Secondary Outcome: Rate of All AEs Per Infusion Categorized by MedDRA Preferred Terms, Seriousness and Severity (G-M).
Description: as for outcome 15
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Number of AEs per infusion
  Gastric Stenosis-non-SAE-Mod | 0.001 | 0
  Gastritis-non-SAE-Mild | 0.001 | 0
  Gastroenteritis-non-SAE-Mild | 0.002 | 0
  Gastroenteritis-non-SAE-Mod | 0.001 | 0
  Gastroenteritis Salmonella-non-SAE-Mod | 0.001 | 0
  Gastroenteritis Viral-non-SAE-Mild | 0.003 | 0.002
  Gastroenteritis Viral-non-SAE-Mod | 0.002 | 0.002
  Gastrointestinal Viral Infection-non-SAE-Mild | 0.001 | 0
  Gastrooesophageal Reflux Disease-non-SAE-Mild | 0.002 | 0
  Gastrooesophageal Reflux Disease-non-SAE-Mod | 0.001 | 0
  Genital Herpes-non-SAE-Mild | 0.001 | 0.003
  Genital Herpes-non-SAE-Mod | 0 | 0.002
  Gingival Erosion-non-SAE-Mild | 0.001 | 0
  Gingivitis-non-SAE-Mild | 0.001 | 0
  Glaucoma-non-SAE-Mod | 0.001 | 0
  Glycosuria-non-SAE-Mild | 0.001 | 0
  Gout-non-SAE-Mod | 0.001 | 0
  Haematochezia-non-SAE-Mild | 0.001 | 0
  Haematospermia-non-SAE-Mild | 0.001 | 0
  Haematuria-non-SAE-Mild | 0.001 | 0.002
  Haemoglobin Decreased-non-SAE-Mild | 0 | 0.002
  Haemolysis-non-SAE-Mild | 0.001 | 0
  Haemorrhoids-non-SAE-Mild | 0.001 | 0
  Haemorrhoids-non-SAE-Mod | 0.001 | 0
  Hand Fracture-non-SAE-Mod | 0.001 | 0
  Headache-non-SAE-Mild | 0.026 | 0.065
  Headache-non-SAE-Mod | 0.004 | 0.003
  Heart Rate Irregular-non-SAE-Mild | 0.001 | 0.002
  Herpes Zoster-non-SAE-Mod | 0.002 | 0
  Hiatus Hernia-non-SAE-Mild | 0.001 | 0
  Hydrocele-non-SAE-Mild | 0.001 | 0
  Hypercapnia-non-SAE-Mild | 0.001 | 0
  Hypercholesterolaemia-non-SAE-Mild | 0.001 | 0
  Hypersensitivity-non-SAE-Mild | 0.001 | 0
  Hypertension-non-SAE-Mild | 0.001 | 0.002
  Hypertension-non-SAE-Mod | 0.004 | 0
  Hypertension-SAE-Mod | 0.001 | 0
  Hypoaesthesia-non-SAE-Mild | 0.001 | 0
  Hypokalaemia-non-SAE-Mild | 0 | 0.003
  Hypothyroidism-non-SAE-Mild | 0 | 0.003
  Hypothyroidism-non-SAE-Mod | 0.001 | 0
  Impetigo-non-SAE-Mild | 0.001 | 0
  Incision Site Pain-non-SAE-Mod | 0.001 | 0
  Increased Upper Airway Secretion-non-SAE-Mild | 0.001 | 0
  Inflammation Of Wound-non-SAE-Mild | 0 | 0.002
  Influenza-non-SAE-Mod | 0.004 | 0.007
  Influenza Like Illness-non-SAE-Mild | 0.002 | 0
  Influenza Like Illness-non-SAE-Mod | 0.001 | 0
  Infusion Site Abscess-non-SAE-Mild | 0.001 | 0
  Infusion Site Bruising-non-SAE-Mild | 0.001 | 0
  Infusion Site Discolouration-non-SAE-Mild | 0.001 | 0
  Infusion Site Discomfort-non-SAE-Mild | 0.005 | 0.003
  Infusion Site Erythema-non-SAE-Mild | 0.014 | 0
  Infusion Site Erythema-non-SAE-Mod | 0.001 | 0
  Infusion Site Induration-non-SAE-Mild | 0.001 | 0
  Infusion Site Mass-non-SAE-Mild | 0.001 | 0
  Infusion Site Oedema-non-SAE-Mild | 0.001 | 0
  Infusion Site Pain-non-SAE-Mild | 0.049 | 0.028
  Infusion Site Pain-non-SAE-Mod | 0.004 | 0.003
  Infusion Site Pruritus-non-SAE-Mild | 0.019 | 0
  Infusion Site Swelling-non-SAE-Mild | 0.002 | 0
  Infusion Site Swelling-non-SAE-Sev | 0.001 | 0
  Injection Site Pain-non-SAE-Mild | 0.002 | 0
  Insomnia-non-SAE-Mild | 0.003 | 0
  Insomnia-non-SAE-Mod | 0 | 0.002
  Intervertebral Disc Degeneration-non-SAE-Mild | 0.001 | 0
  Iron Deficiency Anaemia-non-SAE-Mild | 0.001 | 0
  Irritable Bowel Syndrome-non-SAE-Mod | 0.001 | 0
  Jejunal Stenosis-non-SAE-Mod | 0.001 | 0
  Joint Dislocation-non-SAE-Sev | 0.001 | 0
  Joint Injury-non-SAE-Mild | 0.001 | 0
  Joint Swelling-non-SAE-Mod | 0 | 0.002
  Laceration-non-SAE-Mild | 0 | 0.002
  Ligament Sprain-non-SAE-Mild | 0.001 | 0
  Ligament Sprain-non-SAE-Mod | 0.001 | 0.003
  Limb Discomfort-non-SAE-Mild | 0 | 0.002
  Liver Function Test Abnormal-non-SAE-Mild | 0.001 | 0
  Local Swelling-non-SAE-Mild | 0.002 | 0
  Localised Infection-non-SAE-Mod | 0.001 | 0
  Loss Of Consciousness-non-SAE-Mild | 0 | 0.002
  Lyme Disease-non-SAE-Mild | 0.001 | 0
  Lymph Gland Infection-non-SAE-Mod | 0.001 | 0
  Lymphadenitis-non-SAE-Mod | 0 | 0.002
  Lymphadenitis Bacterial-non-SAE-Mild | 0.001 | 0
  Lymphadenopathy-non-SAE-Mild | 0.003 | 0.003
  Lymphopenia-non-SAE-Mild | 0.001 | 0
  Malaise-non-SAE-Mild | 0.002 | 0.002
  Medical Device Pain-non-SAE-Mild | 0.001 | 0
  Memory Impairment-non-SAE-Mild | 0.001 | 0
  Meniscus Injury-non-SAE-Mild | 0.001 | 0
  Menstrual Disorder-non-SAE-Mod | 0.001 | 0
  Mental Status Changes-SAE-Sev | 0.001 | 0
  Micturition Urgency-non-SAE-Mild | 0 | 0.002
  Middle Ear Effusion-non-SAE-Mild | 0 | 0.002
  Migraine-non-SAE-Mild | 0.003 | 0.003
  Migraine-non-SAE-Mod | 0.003 | 0.008
  Migraine-non-SAE-Sev | 0 | 0.002
  Mitral Valve Incompetence-non-SAE-Mild | 0.001 | 0
  Molluscum Contagiosum-non-SAE-Mild | 0.001 | 0.002
  Mouth Ulceration-non-SAE-Mild | 0 | 0.002
  Mucosal Inflammation-non-SAE-Mild | 0.001 | 0
  Muscle Contractions Involuntary-non-SAE-Mild | 0.001 | 0
  Muscle Spasms-non-SAE-Mild | 0.003 | 0
  Muscle Strain-non-SAE-Mild | 0.001 | 0
  Muscular Weakness-non-SAE-Mild | 0 | 0.002
  Muscular Weakness-non-SAE-Mod | 0.001 | 0
  Musculoskeletal Pain-non-SAE-Mild | 0.003 | 0
  Musculoskeletal Pain-non-SAE-Mod | 0.001 | 0.002
  Myalgia-non-SAE-Mild | 0.016 | 0.010
  Myalgia-non-SAE-Mod | 0.002 | 0.003

19. Secondary Outcome: Rate of All AEs Per Infusion Categorized by MedDRA Preferred Terms, Seriousness and Severity (N-Z).
Description: as for outcome 15
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Number of AEs per infusion
  Nasal Congestion-non-SAE-Mild | 0.007 | 0.008
  Nasal Congestion-non-SAE-Mod | 0.001 | 0
  Nasal Discomfort-non-SAE-Mild | 0.001 | 0
  Nasopharyngitis-non-SAE-Mild | 0.004 | 0.008
  Nasopharyngitis-non-SAE-Mod | 0.001 | 0
  Nausea-non-SAE-Mild | 0.024 | 0.028
  Nausea-non-SAE-Mod | 0.004 | 0.013
  Nephrolithiasis-non-SAE-Mild | 0 | 0.002
  Nerve Compression-non-SAE-Mild | 0 | 0.002
  Neutrophil Count Decreased-non-SAE-Mild | 0 | 0.002
  Ocular Hyperaemia-non-SAE-Mild | 0 | 0.002
  Oedema Peripheral-non-SAE-Mild | 0.003 | 0.008
  Oedema Peripheral-non-SAE-Mod | 0.003 | 0.002
  Oral Candidiasis-non-SAE-Mild | 0.001 | 0
  Oral Herpes-non-SAE-Mild | 0.004 | 0.003
  Oral Pain-non-SAE-Mild | 0 | 0.002
  Oral Pain-non-SAE-Mod | 0 | 0.002
  Orchitis-non-SAE-Mod | 0.001 | 0
  Oropharyngeal Pain-non-SAE-Mild | 0.003 | 0.002
  Osteoarthritis-non-SAE-Mild | 0.001 | 0.002
  Osteoarthritis-non-SAE-Mod | 0.001 | 0
  Osteopenia-non-SAE-Mild | 0.001 | 0
  Osteoporosis-non-SAE-Mild | 0 | 0.002
  Otitis Externa-non-SAE-Mild | 0.001 | 0.002
  Otitis Externa-non-SAE-Mod | 0 | 0.002
  Otitis Media-non-SAE-Mod | 0.001 | 0.002
  Pain-non-SAE-Mild | 0.006 | 0
  Pain In Extremity-non-SAE-Mild | 0.003 | 0.002
  Pain In Extremity-non-SAE-Sev | 0 | 0.002
  Palpitations-non-SAE-Mild | 0.001 | 0
  Panic Attack-non-SAE-Mild | 0 | 0.002
  Papule-non-SAE-Mild | 0.001 | 0
  Paraesthesia-non-SAE-Mild | 0.001 | 0
  Paranasal Cyst-non-SAE-Mild | 0.001 | 0
  Pelvic Pain-non-SAE-Mod | 0.001 | 0
  Pericardial Effusion-non-SAE-Mild | 0.001 | 0
  Perineurial Cyst-non-SAE-Mod | 0.001 | 0
  Periodontal Disease-non-SAE-Mild | 0.001 | 0
  Pharyngitis-non-SAE-Mild | 0.004 | 0.002
  Pharyngitis-non-SAE-Mod | 0 | 0.002
  Pharyngitis Streptococcal-non-SAE-Mild | 0.001 | 0
  Pleural Effusion-non-SAE-Mild | 0.001 | 0
  Pleural Effusion-non-SAE-Mod | 0.001 | 0
  Pneumonia-non-SAE-Mild | 0.001 | 0
  Pneumonia Bacterial-non-SAE-Mod | 0.001 | 0
  Pneumonia Pseudomonas Aeruginosa-SAE-Sev | 0.001 | 0
  Pollakiuria-non-SAE-Mild | 0 | 0.002
  Pollakiuria-non-SAE-Mod | 0.001 | 0
  Polycystic Ovaries-non-SAE-Mild | 0 | 0.002
  Post Procedural Complication-non-SAE-Mod | 0.001 | 0
  Post Procedural Haemorrhage-non-SAE-Mild | 0.001 | 0
  Post Procedural Swelling-non-SAE-Mild | 0.001 | 0
  Procedural Nausea-non-SAE-Mod | 0.001 | 0
  Procedural Pain-non-SAE-Mild | 0 | 0.002
  Procedural Pain-non-SAE-Mod | 0.006 | 0.002
  Proctalgia-non-SAE-Mod | 0.001 | 0
  Productive Cough-non-SAE-Mild | 0.001 | 0
  Protein Urine Present-non-SAE-Mild | 0.001 | 0
  Pruritus-non-SAE-Mild | 0.002 | 0.010
  Pruritus-non-SAE-Mod | 0.001 | 0
  Pruritus Allergic-non-SAE-Mod | 0 | 0.002
  Pruritus Generalised-non-SAE-Mild | 0 | 0.002
  Pulmonary Hypertension-non-SAE-Mild | 0.001 | 0
  Pulmonary Hypertension-non-SAE-Mod | 0.001 | 0
  Pulmonary Vascular Disorder-non-SAE-Mod | 0.001 | 0
  Puncture Site Pain-non-SAE-Mild | 0 | 0.002
  Puncture Site Pain-non-SAE-Mod | 0 | 0.003
  Purpura Senile-non-SAE-Mild | 0 | 0.002
  Pyogenic Granuloma-non-SAE-Mod | 0.001 | 0.002
  Pyrexia-non-SAE-Mild | 0.009 | 0.008
  Pyrexia-non-SAE-Mod | 0.001 | 0
  Pyuria-non-SAE-Mild | 0 | 0.002
  Rales-non-SAE-Mod | 0.001 | 0.002
  Rash-non-SAE-Mild | 0.001 | 0.002
  Rash Generalised-non-SAE-Mild | 0 | 0.002
  Rectal Polyp-non-SAE-Mod | 0.001 | 0
  Red Blood Cells Urine Positive-non-SAE-Mild | 0.001 | 0
  Respiratory Tract Congestion-non-SAE-Mild | 0.001 | 0
  Respiratory Tract Congestion-non-SAE-Mod | 0.001 | 0
  Respiratory Tract Infection-non-SAE-Mild | 0.001 | 0
  Respiratory Tract Infection-non-SAE-Mod | 0.001 | 0
  Restless Legs Syndrome-non-SAE-Mild | 0.001 | 0
  Rhinitis-non-SAE-Mild | 0.001 | 0
  Rhinitis Perennial-non-SAE-Mild | 0.001 | 0
  Rhinorrhoea-non-SAE-Mild | 0.001 | 0.003
  Right Atrial Dilatation-non-SAE-Mild | 0.001 | 0
  Rotator Cuff Syndrome-non-SAE-Mild | 0.001 | 0
  Scab-non-SAE-Mild | 0.001 | 0
  Scar-non-SAE-Mild | 0.001 | 0
  Scoliosis-non-SAE-Mild | 0 | 0.002
  Scratch-non-SAE-Mild | 0.001 | 0
  Scrotal Swelling-non-SAE-Mild | 0.002 | 0
  Seborrhoeic Keratosis-non-SAE-Mod | 0.001 | 0
  Sinus Congestion-non-SAE-Mild | 0.001 | 0.002
  Sinus Headache-non-SAE-Mild | 0.001 | 0
  Sinusitis-non-SAE-Mild | 0.021 | 0.005
  Sinusitis-non-SAE-Mod | 0.018 | 0.022
  Skin Hyperpigmentation-non-SAE-Mild | 0.001 | 0
  Skin Lesion-non-SAE-Mild | 0.001 | 0
  Skin Mass-non-SAE-Mild | 0.001 | 0.002
  Sleep Apnoea Syndrome-non-SAE-Mild | 0.001 | 0
  Slow Speech-non-SAE-Mod | 0.001 | 0
  Solar Lentigo-non-SAE-Mild | 0.001 | 0
  Somnolence-non-SAE-Mild | 0.001 | 0
  Speech Disorder-non-SAE-Mild | 0 | 0.002
  Spermatocele-non-SAE-Mild | 0.001 | 0
  Spinal Compression Fracture-non-SAE-Mod | 0.001 | 0
  Spinal Meningeal Cyst-SAE-Sev | 0.001 | 0
  Spinal Osteoarthritis-non-SAE-Mild | 0.002 | 0
  Squamous Cell Carcinoma-non-SAE-Mod | 0.003 | 0.003
  Stress-non-SAE-Mod | 0.001 | 0
  Suicide Attempt-non-SAE-Sev | 0.001 | 0
  Sunburn-non-SAE-Mild | 0.001 | 0
  Swelling Face-non-SAE-Mod | 0.001 | 0
  Swelling Face-non-SAE-Sev | 0 | 0.002
  Swollen Tongue-non-SAE-Mild | 0.001 | 0
  Synovial Cyst-non-SAE-Mild | 0.001 | 0
  Tachycardia-non-SAE-Mild | 0.003 | 0.002
  Tachycardia-non-SAE-Mod | 0.001 | 0
  Tendon Disorder-non-SAE-Sev | 0.001 | 0
  Tendonitis-non-SAE-Mild | 0.001 | 0
  Tendonitis-non-SAE-Mod | 0.001 | 0
  Testicular Microlithiasis-non-SAE-Mild | 0.001 | 0
  Testicular Pain-non-SAE-Mod | 0.001 | 0
  Thermal Burn-non-SAE-Mild | 0 | 0.002
  Thinking Abnormal-non-SAE-Mod | 0.001 | 0
  Thrombocytopenia-non-SAE-Mild | 0.001 | 0
  Tibia Fracture-non-SAE-Sev | 0.001 | 0
  Tinea Cruris-non-SAE-Mild | 0.001 | 0
  Tinea Infection-non-SAE-Mild | 0.001 | 0
  Tooth Abscess-non-SAE-Mild | 0 | 0.002
  Tooth Abscess-non-SAE-Mod | 0 | 0.002
  Tooth Fracture-non-SAE-Mod | 0.001 | 0
  Tooth Infection-non-SAE-Mild | 0.001 | 0
  Tooth Infection-non-SAE-Mod | 0.001 | 0
  Toothache-non-SAE-Mod | 0 | 0.002
  Toxicity To Various Agents-SAE-Sev | 0.001 | 0
  Tracheal Stenosis-non-SAE-Mild | 0 | 0.002
  Transient Ischaemic Attack-SAE-Mod | 0 | 0.002
  Traumatic Haematoma-non-SAE-Mild | 0.001 | 0
  Tricuspid Valve Incompetence-non-SAE-Mild | 0.001 | 0
  Trigeminal Neuralgia-non-SAE-Mild | 0.001 | 0
  Tympanic Membrane Scarring-non-SAE-Mild | 0.001 | 0
  Type 2 Diabetes Mellitus-non-SAE-Mod | 0.001 | 0
  Upper Limb Fracture-non-SAE-Mod | 0.001 | 0
  Upper Limb Fracture-non-SAE-Sev | 0.001 | 0
  Upper Respiratory Tract Infection-non-SAE-Mild | 0.010 | 0.013
  Upper Respiratory Tract Infection-non-SAE-Mod | 0.008 | 0.003
  Upper-Airway Cough Syndrome-non-SAE-Mild | 0.001 | 0.002
  Urethritis-non-SAE-Mild | 0.001 | 0
  Urinary Tract Infection-non-SAE-Mild | 0.003 | 0.007
  Urinary Tract Infection-non-SAE-Mod | 0.004 | 0.003
  Urticaria-non-SAE-Mild | 0 | 0.003
  Uterine Polyp-non-SAE-Mod | 0.001 | 0
  Vaginal Prolapse-SAE-Mod | 0.001 | 0
  Vaginitis Bacterial-non-SAE-Mild | 0.001 | 0
  Varicose Vein-non-SAE-Mild | 0.001 | 0
  Vasomotor Rhinitis-non-SAE-Mild | 0.001 | 0
  Vein Pain-non-SAE-Mild | 0 | 0.002
  Ventricular Hypokinesia-non-SAE-Mild | 0.001 | 0
  Vessel Puncture Site Bruise-non-SAE-Mild | 0.001 | 0
  Viral Infection-non-SAE-Mild | 0.002 | 0
  Viral Infection-non-SAE-Mod | 0 | 0.002
  Viral Pharyngitis-non-SAE-Mild | 0.001 | 0
  Viral Pharyngitis-non-SAE-Mod | 0 | 0.002
  Viral Rash-non-SAE-Mod | 0.001 | 0
  Viral Upper Respiratory Tract Inf.-non-SAE-Mild | 0.018 | 0.008
  Viral Upper Respiratory Tract Inf-non-SAE-Mod | 0.001 | 0.002
  Vision Blurred-non-SAE-Mild | 0.001 | 0
  Vitamin B12 Deficiency-non-SAE-Mild | 0.001 | 0
  Vitamin D Decreased-non-SAE-Mild | 0 | 0.002
  Vitamin D Deficiency-non-SAE-Mild | 0.001 | 0
  Vitamin D Deficiency-non-SAE-Mod | 0.001 | 0
  Vomiting-non-SAE-Mild | 0.008 | 0.003
  Vomiting-non-SAE-Mod | 0.003 | 0.003
  Vulvar Dysplasia-non-SAE-Mild | 0.001 | 0
  Vulvovaginal Candidiasis-non-SAE-Mild | 0.001 | 0
  Vulvovaginal Mycotic Infection-non-SAE-Mild | 0.003 | 0.002
  Vulvovaginal Mycotic Infection-non-SAE-Mod | 0.001 | 0
  Wheezing-non-SAE-Mod | 0.001 | 0
  Wisdom Teeth Removal-non-SAE-Mild | 0.001 | 0
  Wisdom Teeth Removal-non-SAE-Sev | 0.001 | 0
  Wound-non-SAE-Mild | 0 | 0.002
  Wrist Fracture-non-SAE-Mod | 0 | 0.002
  Xeroderma-non-SAE-Mild | 0.001 | 0

20. Secondary Outcome: Rate of AEs Per Participant (Including and Excluding Infections) Determined by the Investigator to be Related to the Study Drug That Occur at Any Time During the Study ("Related")
Description: Categories presented as adverse event (AE) type : Total, Local, Systemic including infections, Systemic excluding infections, and Severity (Mild, Moderate, Severe, Total). All of these adverse events are non-serious AEs.
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs per participant
  Total AEs, Mild | 4.635 | 2.137
  Total AEs, Moderate | 0.476 | 0.392
  Total AEs, Severe | 0.016 | 0.059
  Total AEs, Total | 5.127 | 2.588
  Local nsAEs, Mild | 2.476 | 0.373
  Local AEs, Moderate | 0.111 | 0
  Local AEs, Severe | 0.016 | 0
  Local AEs, Total | 2.603 | 0.373
  Systemic AEs including infections, Mild | 2.159 | 1.765
  Systemic AEs including infections, Moderate | 0.365 | 0.392
  Systemic AEs including infections, Severe | 0 | 0.059
  Systemic AEs including infections, Total | 2.524 | 2.216
  Systemic AEs excluding infections, Mild | 2.159 | 1.765
  Systemic AEs excluding infections, Moderate | 0.365 | 0.392
  Systemic AEs excluding infections, Severe | 0 | 0.059
  Systemic AEs excluding infections, Total | 2.524 | 2.216

21. Secondary Outcome: Rate of AEs Per Infusion (Including and Excluding Infections) Determined by the Investigator to be Related to the Study Drug That Occur at Any Time During the Study ("Related")
Description: as for outcome 20
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Number of AEs per infusion
  Total AEs, Mild | 0.183 | 0.182
  Total AEs, Moderate | 0.019 | 0.033
  Total AEs, Severe | 0.001 | 0.005
  Total AEs, Total | 0.202 | 0.221
  Local AEs, Mild | 0.098 | 0.032
  Local AEs, Moderate | 0.004 | 0
  Local AEs, Severe | 0.001 | 0
  Local AEs, Total | 0.103 | 0.032
  Systemic AEs including infections, Mild | 0.085 | 0.151
  Systemic AEs including infections, Moderate | 0.014 | 0.033
  Systemic AEs including infections, Severe | 0 | 0.005
  Systemic AEs including infections, Total | 0.099 | 0.189
  Systemic AEs excluding infections, Mild | 0.085 | 0.151
  Systemic AEs excluding infections, Moderate | 0.014 | 0.033
  Systemic AEs excluding infections, Severe | 0 | 0.005
  Systemic AEs excluding infections, Total | 0.099 | 0.189

22. Secondary Outcome: Rate of AEs Per Participant (Including and Excluding Infections) Temporarily Associated With the Infusion
Description: Categories presented as adverse event (AE) type : Total, Local, Systemic including infections, Systemic excluding infections, Seriousness: Serious AE (SAE), non-serious AE (nsAE) and Severity (Mild, Moderate, Severe, Total). All of these adverse events are non-serious AEs.
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per participant
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number of AEs per participant
  Total, nsAE, Mild | 5.921 | 2.275
  Total, nsAE, Moderate | 1.111 | 0.647
  Total, nsAE, Severe | 0.032 | 0.059
  Total nsAE, Total | 7.063 | 2.980
  Total, SAE, Moderate | 0.016 | 0
  Total, SAE, Severe | 0.016 | 0
  Total, SAE, Total | 0.032 | 0
  Local, nsAE, Mild | 2.492 | 0.353
  Local, nsAE, Moderate | 0.111 | 0.039
  Local, nsAE, Severe | 0.016 | 0
  Local, nsAE, Total | 2.619 | 0.392
  Systemic including infections, nsAE, Mild | 3.429 | 1.922
  Systemic including infections, nsAE, Moderate | 1.000 | 0.608
  Systemic including infections, nsAE, Severe | 0.016 | 0.059
  Systemic including infections, nsAE, Total | 4.444 | 2.588
  Systemic including infections, SAE, Moderate | 0.016 | 0
  Systemic including infections, SAE, Severe | 0.016 | 0
  Systemic including infections, SAE, Total | 0.032 | 0
  Systemic excluding infections, nsAE, Mild | 3.111 | 1.922
  Systemic excluding infections, nsAE, Moderate | 0.873 | 0.608
  Systemic excluding infections, nsAE, Severe | 0.016 | 0.059
  Systemic excluding infections, nsAE, Total | 4.000 | 2.588
  Systemic excluding infections, SAE, Moderate | 0.016 | 0
  Systemic excluding infections, SAE, Severe | 0.016 | 0
  Systemic excluding infections, SAE, Total | 0.032 | 0

23. Secondary Outcome: Rate of AEs Per Infusion (Including and Excluding Infections) Temporarily Associated With the Infusion
Description: Categories presented as adverse event (AE) type : Total, Local, Systemic including infections, Systemic excluding infections, Seriousness: Serious AE (SAE), non-serious AE (non-SAE) and Severity (Mild, Moderate, Severe, Total). All of these adverse events are non-serious AEs.
Time Frame: as for outcome 4
Population: Safety Analysis Data Set
Measure: Number; unit: Number of AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 63 | 51
Number analyzed (Infusions) | 1600 | 598
Number of AEs per infusion
  Total, non-SAE, Mild | 0.233 | 0.194
  Total, non-SAE, Moderate | 0.044 | 0.055
  Total, non-SAE, Severe | 0.001 | 0.005
  Total non-SAE, Total | 0.278 | 0.254
  Total, SAE, Moderate | 0.001 | 0
  Total, SAE, Severe | 0.001 | 0
  Total, SAE, Total | 0.001 | 0
  Local, non-SAE, Mild | 0.098 | 0.030
  Local, non-SAE, Moderate | 0.004 | 0.003
  Local, non-SAE, Severe | 0.001 | 0
  Local, non-SAE, Total | 0.103 | 0.033
  Systemic including infections, non-SAE, Mild | 0.135 | 0.164
  Systemic including infections, non-SAE, Moderate | 0.039 | 0.052
  Systemic including infections, non-SAE, Severe | 0.001 | 0.005
  Systemic including infections, non-SAE, Total | 0.175 | 0.221
  Systemic including infections, SAE, Moderate | 0.001 | 0
  Systemic including infections, SAE, Severe | 0.001 | 0
  Systemic including infections, SAE, Total | 0.001 | 0
  Systemic excluding infections, non-SAE, Mild | 0.123 | 0.156
  Systemic excluding infections, non-SAE, Moderate | 0.034 | 0.043
  Systemic excluding infections, non-SAE, Severe | 0.001 | 0.005
  Systemic excluding infections, non-SAE, Total | 0.158 | 0.204
  Systemic excluding infections, SAE, Moderate | 0.001 | 0
  Systemic excluding infections, SAE, Severe | 0.001 | 0
  Systemic excluding infections, SAE, Total | 0.001 | 0

24. Secondary Outcome: Percentage of Infusions Associated With One or More Local AEs (Including and Excluding Infections), at Any Time During the Study
Time Frame: as for outcome 4
Population: Safety Analysis Set
Measure: Number; unit: Percentage of infusions
Units Other Than Participants: Infusions
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Number analyzed (Participants) | 66 | 48
Number analyzed (Infusions) | 1600 | 598
Percentage of infusions
  Including Infections | 8.8 | 3.7
  Excluding Infections | 8.7 | 3.7

ADVERSE EVENTS:
Arm/Group | IGSC, 10% - rHuPH20 | Safety Follow-up - IGSC, 10% or IGIV, 10% Only
Serious Adverse Events (participants affected / at risk) | 9/63 | 3/51
Other Adverse Events (participants affected / at risk) | 60/63 | 45/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGSC, 10% - rHuPH20 (N=63) | Safety Follow-up - IGSC, 10% or IGIV, 10% Only (N=51)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cryptosporidiosis Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Pseudomonas Aeruginosa (Infections and infestations) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Meningeal Cyst (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Adhesiolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGSC, 10% - rHuPH20 (N=63) | Safety Follow-up - IGSC, 10% or IGIV, 10% Only (N=51)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (5) | 1 (2)
Tachycardia (Cardiac disorders) | 5 (6) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (7) | 2 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (8) | 0 (0)
Apthous Stomatitis (Gastrointestinal disorders) | 4 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (19) | 3 (5)
Gastrooesophageal Reflux (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (46) | 4 (25)
Vomiting (Gastrointestinal disorders) | 13 (17) | 2 (4)
Asthenia (General disorders) | 4 (16) | 1 (1)
Fatigue (General disorders) | 11 (27) | 5 (23)
Infusion Site Discomfort (General disorders) | 5 (8) | 1 (2)
Infusion Site Erythema (General disorders) | 12 (23) | 0 (0)
Infusion site Pain (General disorders) | 16 (84) | 2 (19)
Infusion Site Pruritus (General disorders) | 6 (31) | 0 (0)
Oedema Peripheral (General disorders) | 3 (8) | 6 (6)
Pain (General disorders) | 4 (9) | 0 (0)
Pyrexia (General disorders) | 10 (16) | 4 (5)
Bronchitis (Infections and infestations) | 14 (22) | 6 (7)
Cellulitis (Infections and infestations) | 4 (4) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 5 (8) | 2 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 7 (7) | 2 (2)
Influenza (Infections and infestations) | 5 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (8) | 1 (5)
Oral Herpes (Infections and infestations) | 5 (7) | 2 (2)
Pharyngitis (Infections and infestations) | 5 (6) | 2 (2)
Sinusitis (Infections and infestations) | 25 (63) | 11 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (29) | 9 (10)
Urinary Tract Infection (Infections and infestations) | 5 (10) | 5 (6)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 16 (30) | 3 (6)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 8 (9) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 8 (9) | 2 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (28) | 3 (8)
Dizziness (Nervous system disorders) | 6 (11) | 1 (1)
Headache (Nervous system disorders) | 24 (47) | 10 (41)
Migraine (Nervous system disorders) | 6 (9) | 4 (8)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 (32) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 3 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 2 (5)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dermititis Contact (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (6)
Hypertension (Vascular disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxalta requires a review of results communications (e.g., for confidential information) ≥45 days prior to submission or communication. Baxalta may request an additional delay of ≤60 days eg, for intellectual property protection.